# STATISTICAL ANALYSIS PLAN PHASE 2

#### **DATE OF PLAN:**

17 JAN 2012

#### **BASED ON:**

Protocol Amendment 1 on 17 August 2011

*CRF Study Design Version 2.1 on 24 October 2011 (by Central Designer™)* 

#### **STUDY DRUG:**

RUXOLITINIB PHOSPHATE TABLETS / INC 18424

#### PROTOCOL NUMBER:

258

#### **STUDY TITLE:**

AN OPEN LABEL ASSESSMENT OF SAFETY AND EFFICACY OF RUXOLITINIB (INCB018424) IN SUBJECTS WITH PRIMARY MYELOFIBROSIS, POST ESSENTIAL THROMBOCYTHEMIA-MYELOFIBROSIS AND POST POLYCYTHEMIA VERA-MYELOFIBROSIS WHO HAVE PLATELET COUNTS OF 50 x 10<sup>9</sup>/L TO 100 x 10<sup>9</sup>/L

#### **SPONSOR:**

Incyte Corporation
Route 141 & Henry Clay Road
Building E336
Wilmington, DE 19880 United States

This study is being conducted in compliance with good clinical practice, including the archiving of essential documents.

## **Statistical Analysis Plan Approval**

| SAP ID: | INCB 18424-258 SAP |
|--------------------------|----------------------------------|
| SAP Version ID: | Version 1 – Final |
| Submitter | , PhD |
| Date Submitted: | 13 January 2012 |
| <b>Protocol Version:</b> | 17 August 2011 (Amendment 1) |
| CRF Approval Date: | |
| Approval of initial | SAP Approval of Amendment of SAP |

#### NOTE:

- 1) An amendment made prior to the release of unblinded data (eg, treatment assignment received by each subject) for a blinded study or database release for an open-labeled study must be included in an updated SAP.
- 2) An amendment made to the statistical analyses defined in the SAP which occurs after unblinding or database release must be documented in the final Clinical Study Report.
- 3) The approvers must ensure that all relevant functions are in agreement with the final SAP.

This document has been reviewed and accepted by:

| 17 | 2012 |
| Date |

# **TABLE OF CONTENTS**

| 1. | LIST OF ABBREVIATIONS | 6 |
|----------|-------------------------------------------|----|
| 2. | INTRODUCTION | 9 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 10 |
| 3.1. | Study Objectives and Endpoints | 10 |
| 3.1.1. | Study Objectives | 10 |
| 3.1.2. | Study Endpoints | 10 |
| 3.1.2.1. | Co-Primary Endpoints | 10 |
| 3.1.2.2. | Safety Endpoint(s) | 10 |
| 3.1.2.3. | Secondary Endpoints | 11 |
| | | 11 |
| 3.2. | Statistical Hypotheses | 11 |
| 4. | STUDY DESIGN | 12 |
| 4.1. | Overall Description | 12 |
| 4.2. | Scheduled Visits | 13 |
| 4.3. | Sample Size Considerations | 16 |
| 5. | DATA HANDLING DEFINITIONS AND CONVENTIONS | 18 |
| 5.1. | Scheduled Analyses | 18 |
| 5.1.1. | First DMC Data Review Meeting | 18 |
| 5.1.2. | Second DMC Data Review Meeting | 18 |
| 5.2. | Treatment Groups | 19 |
| 5.3. | Analysis Populations | 19 |
| 5.3.1. | Safety Population | 19 |
| 5.3.2. | Intent-to-Treat Population | 19 |
| 5.3.3. | Per-Protocol Population | 19 |
| | | 19 |
| 5.4. | Statistical Methodology | 19 |
| 5.4.1. | General Methodology | 19 |
| 5.4.2. | Control of Type I Error | 20 |
| 5.5. | Baseline Values | 20 |
| 5.6. | Day 1, Study Day, and Study Time Points | 20 |
| 5.7. | Concomitant Medications and Partial Dates | 21 |

| 5.8. | Adverse Events and Missing Data | 22 |
|----------|------------------------------------------------------------|----|
| 5.9. | Variable Definitions and/or Derivation Rules | 23 |
| 5.9.1. | Spleen Volume Value at Week 24 | 23 |
| 5.9.2. | Total Symptom Score | 23 |
| 5.9.2.1. | Daily Total Symptom Score | 23 |
| 5.9.2.2. | Baseline Total Symptom Score | 23 |
| 5.9.2.3. | Total Symptom Score at Weeks 4, 8, 12, 16, 20, and 24 | 24 |
| 5.9.3. | Dosing Level and Compliance | 24 |
| 5.9.3.1. | Final Titrated Dose Level | 24 |
| 5.9.3.2. | Last Average Daily Dose Level During the Treatment Period | 24 |
| 5.9.3.3. | Study Drug Compliance | 25 |
| 5.9.3.4. | Last Dose Level Prior to an Adverse Event. | 25 |
| 5.9.4. | Blood Transfusion Independence at Baseline | 25 |
| 5.9.5. | Blood Transfusion Independence at Post-Baseline | 26 |
| 5.9.6. | Derivation of Per-protocol Population | 26 |
| 6. | BASELINE, EXPOSURE, AND DISPOSITION VARIABLES AND ANALYSES | 27 |
| 6.1. | Baseline and Demographics | 27 |
| 6.2. | Disposition and Enrollment | 27 |
| 6.3. | Protocol Deviations | 27 |
| 6.4. | Exposure | 27 |
| 6.5. | Study Medication Compliance | 27 |
| 6.6. | Medical History | 27 |
| 6.7. | Concomitant Medication | 28 |
| 6.8. | Blood Transfusion Dependency | 28 |
| 7. | EFFICACY ANALYSES | 29 |
| 7.1. | Primary Efficacy Endpoints | 29 |
| 7.2. | Secondary Endpoint(s) and Analyses | 29 |
| | | 30 |
| 8. | SAFETY ANALYSES | 31 |
| 8.1. | Adverse Events | 31 |
| 8.2. | Laboratory Values | 32 |
| 8.3. | Vital Signs | 33 |

| 8.4. | Electrocardiograms | 33 |
|---|---|---|
| 9. | CLINICAL PHARMACOLOGY/ | |
| | | 34 |
| 0.2 | Subject Demonstration Clinical Laboratory and Discoss Deleted Westelland | 34 |
| <ul><li>9.2.</li><li>9.3.</li></ul> | Subject Demographic, Clinical Laboratory, and Disease-Related Variables Concomitant Medication | |
| 9.3. | Concomitant iviedication | 34 |
| | | 35 |
| | | 35 |
| 10. | LIST OF PLANNED TABLES, LISTINGS, AND FIGURES | |
| 10.1. | Tables | |
| 10.2. | Figures | |
| 10.3. | Listings | |
| 11. | REFERENCES | |
| 12. | APPENDICES | 42 |
| APPENDI | X A. MEDDRA PREFERRED TERMS INCLUDED IN THE SMQ TO IDENTIFY HEMORRHAGE ADVERSE EVENTS | 43 |
| APPENDI | X B. SHELLS FOR POST-TEXT TABLES | 51 |
| | LIST OF TABLES | |
| Table 1: | List of Abbreviations | 6 |
| Table 2: | List of Assessments | 14 |
| Table 3: | Table of Laboratory Assessments | 15 |
| Table 4: | Windows for Total Symptom Score at Given Study Time Points | 24 |
| Table 5: | Example Shift Summary for Applicable Laboratory Assessments | 33 |
| Table 6: | High and Low Threshold Values for Alert Vital Sign Observations | 33 |
| | LIST OF FIGURES | |
| Figure 1: | Power and Sample Size Curves for 3 Alternative Hypotheses on the Level of Dose-Effect Correlation | 16 |

# 1. LIST OF ABBREVIATIONS

**Table 1:** List of Abbreviations

| Abbreviation | Term |
|---|---|
| AE | Adverse event |
| ALB | Albumin (G/L) |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| AUC | Area under the concentration-time curve |
| $\mathrm{AUC}_{(0-\infty)}$ | AUC from time zero (pre-dose) extrapolated to infinite time |
| $\mathrm{AUC}_{(0\text{-}	au)}$ | AUC from time zero (pre-dose) to time of last observed quantifiable concentration within a subject across all treatments |
| BLQ | Below limit of quantification |
| BMI | Body mass index |
| bid. | Twice daily |
| BP | Blood pressure |
| bpm | Beats per minute |
| BUN | Blood urea nitrogen |
| °C | Degrees Celsius |
| Ca | Calcium |
| Cl | Chloride |
| CLr | Renal clearance |
| C <sub>max</sub> | Maximum observed concentration |
| CRF | Case report form |
| CSR | Clinical study report |
| Ct | Last observed quantifiable concentration |
| DBP | Diastolic blood pressure |
| DL | Deciliter |
| DOB | Date of birth |
| ECG | Electrocardiogram |
| °F | Degrees fahrenheit |
| GCP | Good Clinical Practices |

**Table 1:** List of Abbreviations (Continued)

| Abbreviation | Term |
|-------------------|----------------------------------------------------------|
| GGT | Gamma-glutamyl transferase |
| HGB | Hemoglobin |
| In | Inches |
| IP | Investigational product |
| IRB | Institutional Review Board |
| ITT | Intent-to-treat population |
| IU | International units |
| K | Potassium |
| $\lambda_{\rm z}$ | Terminal phase rate constant |
| LDH | Lactate dehydrogenase |
| LFTs | Liver function tests |
| LLN | Lower limit of normal |
| MedDRA | Medical Dictionary for Regulatory Activities Terminology |
| mg | Milligrams |
| mL | Milliliter |
| mmHg | Millimeters of mercury |
| msec | Milliseconds |
| Na | Sodium |
| ng | Nanograms |
| PET-MF | Post Essential Thrombocythemia-Myelofibrosis |
| PMF | Primary Myelofibrosis |
| PP | Per-protocol population |
| PPV-MF | Post Polycythemia Vera-Myelofibrosis |
| RBC | Red blood cell count |
| SAE | Serious adverse event |
| SAS | Statistical Analysis System |
| SBP | Systolic blood pressure |
| SGOT | Serum glutamic oxaloacetic transaminase |
| SGPT | Serum glutamic pyruvic transaminase |

**Table 1:** List of Abbreviations (Continued)

| Abbreviation | Term |
|------------------|----------------------------------------|
| t <sub>1/2</sub> | Terminal phase half-life |
| t <sub>max</sub> | Time of occurrence of C <sub>max</sub> |
| TIBC | Total iron binding capacity |
| UIBC | Unsaturated iron-binding capacity |
| ULN | Upper limit of normal |
| WBC | White blood cell count |
| WHO | World Health Organization |

#### 2. INTRODUCTION

The purpose of this document is to provide a detailed statistical analysis plan (SAP) for the data collected during the conduct of the study protocol (entitled "An open label assessment of safety and efficacy of ruxolitinib (INCB018424) in subjects with primary myelofibrosis (PMF), post essential thrombocythemia-myelofibrosis (PET-MF) and post polycythemia vera-myelofibrosis (PPV-MF) who have platelet counts of 50 x 10<sup>9</sup>/L to 100 x 10<sup>9</sup>/L", Amendment 1 dated 17 August 2011) which will be analyzed, summarized, and presented in the clinical study report (CSR). The case report form (CRF) version covered by this SAP is Study Design Version 1.6 (dated 28 July 2011, generated by Central Designer<sup>TM</sup>).

Section 4 of the protocol provides a detailed description of the investigational product, target patient population, the rationale for doses to be examined, and the potential risks and benefits of ruxolitinib (INCB018424).

#### 3. STUDY OBJECTIVES AND ENDPOINTS

## 3.1. Study Objectives and Endpoints

#### 3.1.1. Study Objectives

#### **Primary Objectives:**

- To determine the effects of ruxolitinib on spleen volume and symptom burden in patients with PMF, PPV-MF, and PET-MF who have a baseline platelet count of 50 x 10<sup>9</sup>/L to 100 x 10<sup>9</sup>/L.
- To determine the safety and tolerability of ruxolitinib in subjects with PMF, PPV-MF, and PET-MF who have a baseline platelet count of  $50 \times 10^9$ /L to  $100 \times 10^9$ /L.

#### **Secondary Objective:**

• To determine an appropriate dosing strategy for subjects with low platelets.

#### 3.1.2. Study Endpoints

## 3.1.2.1. Co-Primary Endpoints

- Correlation of percent change from baseline in spleen volume at Week 24 versus final titrated dose.
- Correlation of percent change from baseline in total symptom score as measured by the modified MFSAF v2.0 diary at Week 24 versus final titrated dose.

#### 3.1.2.2. Safety Endpoint(s)

- Safety and tolerability will be assessed by monitoring the frequency, duration, and severity of adverse events (AEs), performing physical examinations, collecting vital signs, collecting laboratory data for hematology, serum chemistry, coagulation parameters, and urinalysis. In addition, analyses will include:
  - Proportion of subjects with new onset Grade 4 thrombocytopenia events as assessed by CTCAE v4.03;
  - Proportion of subjects with new onset Grade 2 or higher hemorrhage as assessed by CTCAE v4.03.

#### 3.1.2.3. Secondary Endpoints

- Percent change from baseline in spleen volume at Week 24.
- Percent change from baseline in total symptom score as measured by the modified MFSAF v2.0 diary at Week 24.
- Proportion of subjects with ≥ 35% reduction from baseline in spleen volume at Week 24.
- Proportion of subjects with ≥ 10% reduction from baseline in spleen volume at Week 24.
- Proportion of subjects with  $\geq$  50% improvement from baseline in total symptom score as measured by the modified MFSAF v2.0 diary at Week 24.
- Change and percentage change from baseline in spleen length as measured by palpation at each visit where the parameter is assessed.



# 3.2. Statistical Hypotheses

The null hypothesis is that the correlation between percent change in spleen volume or total symptom score and final titrated dose is zero. The alternative hypothesis is that the correlation is not zero.

#### 4. STUDY DESIGN

## 4.1. Overall Description

This is an open label study of 24 weeks duration of ruxolitinib in subjects with PMF, PPV-MF, and PET-MF. The study is comprised of 4 phases (see protocol Section 7.1, Overall Study Design):

**Screening:** up to 21 days. **Baseline:** exactly 7 days.

**Treatment Phase:** 24 weeks. For subjects receiving benefit from treatment, further participation may continue up to the time of commercial availability of ruxolitinib.

**Follow-up Phase:** 30 to 37 days after the last dose of ruxolitinib is taken.

All subjects will begin dosing at 5 mg bid ruxolitinib. Doses should be taken morning and evening, approximately 12 hours apart, and without regard to food.

Doses of ruxolitinib may be increased in 5 mg qd increments up to 10 mg bid starting at the Week 4 visit and at subsequent study visits (no more than every 4 weeks) if subjects meet prespecified criteria (refer to protocol Section 8.6, Dose Adjustments).

Doses may not exceed 10 mg bid except in subjects who continue to meet the dose escalation criteria (see Protocol, Section 8.6, Dose Adjustments), and who have, in addition, a PGIC score of minimally worse, much worse, or very much worse while receiving 10 mg bid. Such subjects may continue dose escalation to a maximum dose of 15 mg bid.

Doses may never exceed 15 mg bid, and no dose increases may occur after Week 16.

Subjects will be required to decrease the dose for platelet count  $< 35 \times 10^9/L$ , and to hold administration for platelet count  $< 25 \times 10^9/L$ . Subjects will have the option to restart or re-escalate the dose with improving platelet count.

Subjects will be required to interrupt administration for any Grade 2 or higher hemorrhage events. Subjects will be able to restart ruxolitinib administration with resolution of Grade 2 events; restart after a second event requires review and discussion of pertinent data with the sponsor. Restarts of ruxolitinib will only be permitted in some cases of Grade 3 and 4 events, after review and discussion of pertinent data with the sponsor.

Sites will provide information on incidents of Grade 4 thrombocytopenia and Grade 3 and Grade 4 hemorrhage events via FAX to the sponsor within 24 hours of learning of the event. The overall incidence of these events will be continuously monitored by the sponsor, and with ongoing data review, could result in a temporary hold for further enrollment, a reduction in the maximum allowable dose for subjects in the study, or a protocol amendment to modify dose titration rules (see protocol Section 11.7, Study Safety Monitoring).

# 4.2. Scheduled Visits

Table 2 (source: protocol Table 3) and Table 3 (source: protocol Table 4) on the next pages provide detailed study visits and measurements of safety and efficacy variables defined for this study.

Table 2: List of Assessments

| Table 2: List o | 1 Assessme<br> Screening | Baseline | Day | Weeks 1,2, | Week | Week | Week | Week | Week | Week | Extension | End of | Follow-Up 30- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 1 | 3,5,6,7,10, 14,<br>18, 28 and q4<br>weeks<br>thereafter | 4 | 8 | 12 | 16 | 20 | 24 | Phase Visits<br>(q12 weeks<br>after Week 24) | Treatment or<br>Early<br>Termination<br>Visit (EOT) | 37 days after<br>last dose of<br>ruxolitinib or<br>EOT visit |
| Evaluation/window | Day -28 to | Day -7 to | Day | ± 3 | ± 5 | ± 5 | ± 5 | ± 5 | ± 5 | ± 5 | ± 5 days | ± 5 days | |
| A serious C. Lineat NI serious | -8 | -1 | 1 | days | days | days | days | days | days | days | | | |
| Assign Subject Number | X<br>X | 37 | | | | | | | | | | | |
| Informed consent /<br>Eligibility Criteria | | X | | | | | | | | | | | |
| Prior Medical & medication history | X | X | | | | | | | | | | | |
| Concomitant medication review | | X | X | | X | X | X | X | X | X | X | X | X |
| Transfusion history/status | X | X | | | X | X | X | X | X | X | X | X | X |
| Discontinue prior MF therapies | X | | | | | | | | | | | | |
| Screening Symptom Form | X | | | | | | | | | | | | |
| Record AEs | X | X | X | | X | X | X | X | X | X | X | X | X |
| Physical examination | X | X | | | | | X | | | X | X | X | X |
| Spleen Palpation | X | X | | | X | X | X | X | X | X | X | X | X |
| Vital Signs | X | X | | | X | X | X | X | X | X | X | X | X |
| 12-lead ECG | X | | | | | | | | | | | | |
| BM biopsy | X | X <sup>a</sup> | | | | | | | | | | | |
| MRI of upper and lower abdomen and pelvis | | X | | | | | | | | X | | | |
| Modified MFSAF v2.0 | | | Diary | y is completed each | evening f | rom Day | -7 to the V | Veek 24 v | visit | | | | |
| Dispense and/or Bring<br>MFSAF v2.0 diary to visit | | X | X | | X | X | X | X | X | X | | | |
| PGIC <sup>b</sup> | | | | | X | X | X | X | X | X | X | X | |
| ECOG status | X | X | | | X | X | X | | | X | X | X | |
| Dispense reminder card | | X | X | | X | X | X | X | X | X | X | | |
| Contact IVRS | X | | X | | X | X | X | X | X | X | X | X | |
| Administer study drug during visit | | | X | | X | | | | | | | | |
| Dispense study drug | | | X | | X | X | X | X | X | X | X | | |
| Drug accountability assessment | | | | | X | X | X | X | X | X | X | X | |

<sup>&</sup>lt;sup>a</sup> If not completed at Screening visit, and biopsy in prior 2 months is not available.

<sup>b</sup> PGIC = Patient Global Impression of Change (protocol Appendix V).

**Table 3:** Table of Laboratory Assessments

| | Screening | Baseline | Day<br>1 | Weeks 1,2,<br>3,5,6,7,10,<br>14, 18, 28<br>and q 4<br>weeks<br>thereafter | Week<br>4 | Week<br>8 | Week<br>12 | Week<br>16 | Week<br>20 | Week<br>24 | Extension<br>Phase Visits<br>(q12 weeks<br>after Week 24) | End of Treatment or Early Termination Visit (EOT) | Follow-Up<br>30 to 37 days<br>after last dose<br>of ruxolitinib<br>or EOT visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Assessment | Day -28 to | Day -7 to | Day | ± 3 | ± 5 | ± 5 | ± 5 | ± 5 | ± 5 | ± 5 days | ± 5 days | ± 5 days | |
| | -8 | -1 | 1 | days | days | days | days | days | days | | | | |
| Serum Chemistry | X | X | | | X | X | X | X | X | X | X | X | X |
| Hematology | X | X | | X | X | X | X | X | X | X | X | X | X |
| Coagulation panel | X | X | | | | | X | | | X | X | X | X |
| Lipid Panel | | X | | | X | | X | | | X | X | X | X |
| Serum Pregnancy Test <sup>a</sup> | X | | | | | | | | | | | | X |
| Urine Pregnancy Test <sup>a</sup> | | X | | | X | X | X | X | X | X | X | X | |
| Serology for HIV,<br>HBV, HCV | X | | | | | | | | | | | | |

| Urinalysis | X | X | X | X | X |
|------------|---|---|---|---|---|

<sup>&</sup>lt;sup>a</sup> Women of childbearing potential only.

## 4.3. Sample Size Considerations

Approximately 150 subjects will be enrolled in order to assess (on the efficacy side) the dose-effect correlation (between percent changes from baseline in spleen volume/total symptom score at Week 24 and final titrated dose level). Using an alpha of 5% (2-sided), this sample size gives a power of 96% to reject the null hypothesis of no dose-effect correlation if the true correlation is 0.30. The power is 87% if the true correlation is 0.25, and the power is 69% if the true correlation is 0.20. These calculations are based on Cohen 1988, Formula 12.3.4. SAS procedure POWER is used and the power curves are displayed in Figure 1.

Figure 1: Power and Sample Size Curves for 3 Alternative Hypotheses on the Level of Dose-Effect Correlation



It is noted that the above sample size calculation is based on the rationale that the first primary endpoint (correlation between percent change from baseline in spleen volume at Week 24 by the final titrated dose) is powered following the procedure of the sequential test used for this study (see Section 5.4.2). At the given sample size, power can also be assessed for the second co-primary endpoint (correlation between percent change from baseline in total symptom score at Week 24 by the final titrated dose.

In addition, the mean percent change from baseline in spleen volume measured by MRI, and mean percent change from baseline in total symptom score at Week 24 will each be estimated with a 95% confidence interval. With 150 subjects, the half-length of the 95% confidence

Incyte Corporation INCB 18424-258

interval of the change from baseline in spleen volume at Week 24 is approximately 3%. This is based on the Phase 3 study (INCB 18424-351), where the standard deviation of the percent change from baseline in spleen volume at Week 24 was 19%.

17

#### 5. DATA HANDLING DEFINITIONS AND CONVENTIONS

## 5.1. Scheduled Analyses

In addition to the planned final CSR analysis, interim data reviews by the DMC focused on events of thrombocytopenia and hemorrhage on predefined schedules are planned.

- 28 days after 20 subjects have enrolled.
- 28 days after 40 subjects have enrolled.
- Other reviews can be scheduled only if the DMC deems it necessary that additional data would need to be reviewed to assess safety parameters as specified by the protocol.

Since all interim data reviews are focused on safety only, there is no alpha-spend of the final CSR efficacy analysis.

#### **5.1.1.** First DMC Data Review Meeting

When the 20th patient is enrolled, additional screening of subjects will be paused for at least 28 days and up to approximately 42 days. Subjects in screening at that time will be allowed to enroll if they are found to be eligible. During this period, enrolled subjects will be allowed to continue on study per the protocol. At least 28 days from the enrollment of the 20th subject, safety data will be assessed by the DMC and the sponsor. Subjects will be analyzed if they have completed at least 28 days on the study or have discontinued the study because of Grade 4 thrombocytopenia or > Grade 2 hemorrhage. Demographics, baseline characteristics, and dose exposure will be summarized for those subjects. Also AE and laboratory parameters will be analyzed.

#### **5.1.2.** Second DMC Data Review Meeting

At least 28 days from the enrollment of the 40th subject, safety data will be assessed by the DMC and the sponsor. Since the first dose escalation opportunity in the study is at Day 28 and the starting dose for all subjects of 5 mg bid will have been adequately assessed for safety at the first safety review after the enrollment of 20 patients, screening will not be suspended following enrollment of the 40th subject. If safety of the 5 mg bid dose is not clear from this first data review, the DMC and the sponsor may mandate a hold on screening at the review that occurs with enrollment of the 40th subject. Subjects will be analyzed when they have completed at least 28 days on the study or discontinued due to Grade 4 thrombocytopenia or > Grade 2 hemorrhage. Demographics, baseline characteristics, and exposure will be summarized for those subjects. Also AE and laboratory parameters will be analyzed.

More details were described in the protocol Section 11.7, Data Safety Monitoring and the corresponding DMC charter.

## **5.2.** Treatment Groups

Subjects will be summarized as 1 group regardless of dose titration. For certain summaries of AEs by dose received (details can be found in the appendix of table shells), subjects will be grouped into the following categories:  $\leq 5$  mg, > 5 to 10 mg, > 10 to 15 mg, > 15 to 20 mg, > 20 to 25 mg, and > 25 mg based on the final titrated total daily dose (see Section 5.9.3.1).

In addition, for the summary of exposure, final titrated dose groups as defined above may be used as treatment groups and additional efficacy analysis may utilize these dose categories.

# 5.3. Analysis Populations

#### **5.3.1.** Safety Population

All subjects who are enrolled and have taken at least 1 dose of study drug comprise the safety population. The safety population will be used to conduct all safety analyses, including baseline and demographics.

#### **5.3.2.** Intent-to-Treat Population

All subjects who are enrolled and have taken at least 1 dose of study drug constitute the intent-to-treat (ITT) population. All efficacy analyses will be conducted using the ITT population. It is noted that the ITT population is effectively identical to the safety population for this study.

#### **5.3.3.** Per-Protocol Population

The per-protocol (PP) population includes those subjects in the ITT population who are considered to be sufficiently compliant with the protocol. The PP population will be used for certain supportive sensitivity analysis of efficacy and safety. Derivation rules for PP population can be found in Section 5.9.6.



# 5.4. Statistical Methodology

#### 5.4.1. General Methodology

Unless otherwise denoted, SAS® procedures (Version 9 or above) will be employed for the generation of all tables, graphs, and statistical analyses.

Descriptive summaries for continuous

deviation, median, minimum, and maximum. Descriptive summaries for categorical variables will include the number and percentage of subjects in each category.

The Safety Population will be used for all safety analyses, and the ITT population will be used for all efficacy analyses. The primary efficacy analysis will also be repeated by using the PP population.

#### **5.4.2.** Control of Type I Error

All confidence intervals will be 95% and tests will be performed at 2-sided 0.05% level. Because of the exploratory nature of the study analyses, except for tests regarding the coprimary endpoints, no multiplicity adjustment will be performed. To control overall Type I error in testing hypotheses regarding the coprimary endpoints, a sequential testing procedure will be used.

- Step 1 will test the correlation between percent change from baseline in spleen volume at Week 24 and the last titrated dose level, and only if the null hypothesis of no correlation can be rejected, Step 2 will be carried out.
- Step 2 will test the correlation between percent change from baseline in total symptom score at Week 24 and the last titrated dose level. In case Step 1 fails to reject the null hypothesis, the inferential comparison (p-values) of Step 2 will still be generated for descriptive purposes only.

#### 5.5. Baseline Values

A baseline value (for analysis purposes) is the last, non-missing measurement obtained during the screening visit and baseline visit unless otherwise stated, with the exception of laboratory values and the total symptom score. For laboratory assessments, values obtained on Day 1 (see Section 5.6) will be included in deriving baseline as the laboratory values are scheduled to be obtained before on-site administration of study drug. For total symptom scores, different derivation rules will be used (see Section 5.9.2.2).

# 5.6. Day 1, Study Day, and Study Time Points

Day 1 is the date of first dose of study medication.

The study day at a visit/reporting date will be calculated by the visit/reporting Date – Day 1 + 1. This study day will be subtracted by 1 if it is less than or equal to zero, so that a study day of zero will never occur. A study day of -1 indicates 1 day prior to Day 1.

Other study time points will use nominal weeks, such as Weeks 4, 8, 12, etc, according to the Schedules of Assessments (see Table 2 and Table 3), as recorded on the CRF, regardless of the actual time windows these visits fall into, unless otherwise stated. This is especially true for analyses such as laboratory values and vital sign values where by-study-week summaries are to be generated, as well as for spleen palpation length over time summaries.

Exceptions to the statements about study time points described above include (but are not limited to) spleen volume at Week 24 (see Section 5.9.1), total symptom score at several major study time points (see Section 5.6), and final titrated dose level (see Section 5.9.3.1).

Another exception is related to spleen palpation length analysis. Per study CRF design, if a subject's EOT Visit coincides with a scheduled visit, then in database, only EOT Visit data will be available. So when a subject has spleen palpation length data collected on an "EOT Visit" (or End of Extension Phase Visit, as appropriate and if applicable), an effort will be made to see if the data actually falls into a scheduled visit, such as Weeks 4, 8, 12, 16, 20, 24 (treatment phase), 36, 48, 60, etc (extension phase) by using the window of Week of scheduled visit\*7 ± 5 days.

Following the situation described above, if EOT data contain spleen volume measurements and the situation is not resolved by the time of database lock, then similar effort will be made by treating spleen volume data labeled from "EOT Visit" as data collected from unscheduled visit. See Section 5.9.1 for how spleen volume data from unscheduled visits will be used in the analysis.

The situation described above is not an issue of importance to other variables such as laboratory values, since in analyses by time point, "EOT" will be one of the time points to be displayed.

#### 5.7. Concomitant Medications and Partial Dates

Prior medication is defined as any non-study medication started prior to the date of first study drug administration.

Concomitant medication is defined as any non-study medication that is:

- Started before the date of first study drug administration and is ongoing throughout the study or ends on/after the date of first study drug administration;
- Started on/after the date of first study drug administration and is ongoing or ends during the course of study medication.

A prior medication could also be classified as "both prior and concomitant medication" if the end date is on or after first dose of study medication. In the listing, it will be indicated whether or not a medication is prior-only, concomitant-only, or both prior and concomitant medication.

The start/stop dates recorded by the Investigator and his/her research staff in the eCRF will be used to identify when a concomitant medication was taken during the study. Any missing start date must be queried for resolution. Unresolved missing start dates will be handled according to the following order of steps.

- If the date is completely missing, the medication will be considered both prior and concomitant.
- If only the day is missing, and the last day of the month is prior the first dose date on Day 1, then the concomitant medication will be considered as starting prior to Day 1, and the incomplete date will be handled as if it is the last day of the month.
- If only the day is missing, and the first day of the month is after the first dose date on Day 1, then the concomitant medication will be considered as starting after Day 1, and the incomplete date will be handled as if it is the first day of the month.
- If only the day is missing, and the month is equal to the month of the first dose date on Day 1, then the missing day will be handled as if it is the first day of the month.
- If both the month and day are missing, and the last day of the year is prior to the first dosing date on Day 1, then the concomitant medication will be considered as starting before Day 1, and the incomplete date will be handled as if it is the last day of the year. Otherwise, the missing date will be handled as if it is the first day of the year.

# 5.8. Adverse Events and Missing Data

A treatment-emergent adverse event (TEAE) is any AE either reported for the first time or worsening of a pre-existing event after first dose of study medication. Analysis of AEs will be limited to TEAEs, but data listings will include all AEs.

Severity of AEs will be described and graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE). CTCAE v4.03 is used for this protocol. If the toxicity is not included in the CTCAE v4.03 criteria it will be rated on a 1 to 4 scale as follows: mild = 1; moderate = 2; severe = 3; and life-threatening = 4.

An AE will also be assessed by its relationship to study medication as well as by seriousness. These assessments will be directly from data collected on eCRFs and are described in details in the protocol.

Any missing onset date, causality, or severity must be queried for resolution. Unsolved missing values will be handled according to the following rules:

- An unsolved missing causality will be considered treatment related
- An unsolved missing severity will be identified as an unknown severity

- For purposes of analysis, all AEs will be considered TEAEs unless the AE can unequivocally be defined as not treatment emergent. Therefore, an unsolved missing onset date will be considered treatment emergent, with the following examples illustrating exceptions:
  - If the stop/resolution date is before the first dose date on Day 1, then the AE will be considered as not being treatment emergent.
  - If both the month and day are missing, and the last day of the year is before the first dose date on Day 1, then the AE will not be considered treatment emergent.
  - If only the day is missing, and the last day of the month is before the first dose date on Day 1, then the AE will not be considered treatment emergent.
  - If only the day is missing, and the first day of the month is after the first dosing date on Day 1, then the AE will be considered treatment emergent.

#### 5.9. Variable Definitions and/or Derivation Rules

#### 5.9.1. Spleen Volume Value at Week 24

If Week 24 spleen volume value is obtained in the manner of by-schedule visit, it will be used as the analytic value for study analysis regardless of the actual time window it falls into. However, if the only values available are from unscheduled visits, then the last available value within the window of Day 141 to Day 175 (=168 + 7 days) will be used as Week 24 spleen volume analytic value. When spleen volume data are available for both by-schedule and unscheduled visits (within the window), the value from the scheduled visit will be used.

#### **5.9.2.** Total Symptom Score

#### 5.9.2.1. Daily Total Symptom Score

Daily total symptom score is derived as the sum of 6 individual symptom scores (the total score excludes scores for degree of inactivity); this score will be missing if there are any missing individual scores. Observations with an un-resolved missing date will be excluded from analysis.

#### **5.9.2.2.** Baseline Total Symptom Score

Baseline value of total symptom score is derived as the average of the prorated daily total symptom score for the 7 days before the first dose on Day 1 (ie, from Day -7 to Day -1). If  $\geq 4$  daily total symptom score values are missing during this period of time, the baseline total symptom score value is set as missing.

#### 5.9.2.3. Total Symptom Score at Weeks 4, 8, 12, 16, 20, and 24

Week X (where X = 4, 8, 12, 16, 20, and 24) total symptom score is derived as the average of the daily total symptom scores collected from the last 28 consecutive days covering the interval between up to Day (X+n)\*7, where n is 1 for Week 24 and 0 otherwise, and Day (X-4)\*7+1 as presented in Table 4.

Table 4: Windows for Total Symptom Score at Given Study Time Points

| <b>Study Time Point</b> | Window | Note |
|---|---|---|
| Week 4 | Day 1 to Day 28 | |
| Week 8 | Day 29 to Day 56 | |
| Week 12 | Day 57 to Day 84 | |
| Week 16 | Day 85 to Day 112 | |
| Week 20 | Day 113 to Day 140 | |
| Week 24 | Last 28 days of the window from Day 141 to the last day when daily total symptom score value is available and it is ≤ Day 175. | If the last evaluation day is before Day 168-7 = 161 then total symptom score will be set as missing for Week 24. |

Total symptom score for given study time points displayed above will be missing if there are more than 8 values missing in the 28-day window. It should be noted that a score of 0 is not a missing value.

## **5.9.3.** Dosing Level and Compliance

#### **5.9.3.1.** Final Titrated Dose Level

The analytic value of the last titrated dose level will be derived as the average of the total daily dose (excluding periods of dose interruption) during the time interval of Day 141 and Day 168, or the last 28 days of available dosing data (for subjects who discontinued treatment early). All available data points in the time interval will be used for this calculation.

### 5.9.3.2. Last Average Daily Dose Level During the Treatment Period

For subjects who have the analytic value of the last titrated dose level derived, the last average daily dose level during the treatment period will be the same. For subjects who discontinued and do not have last titrated dose level derived, it will be the average of the last 28 days (excluding periods of dose interruption) of treatment. For subjects who discontinued study before Day 28, it is the same as the average daily dose level during the study.

#### 5.9.3.3. Study Drug Compliance

Study drug compliance (%) is calculated as

 $100 \times [\text{total dose taken}]/[\text{total dose prescribed}]$ 

where total dose taken is calculated as before, and total dose prescribed will be based on the dosing prescription as collected through the CRF pages of EX domain. If prescribed dose collected from EX domain is 0, it also indicates a prescribed dose interruption; in addition, dose reduction or increase as recorded in EX domain are all regarded as investigator-mandated prescriptions on study drug for the subjects to follow.

Study drug compliance will be calculated only for the pre-extension phase of 24 weeks. Based on need of exploratory analysis, compliance for other periods may be derived as well.

Because of the eCRF design, other than calculating study drug compliance, data collected on the EX domain of the eCRF will be used as actual study drug administration information in order to carry out other dose-response type analyses, such as AEs by the dose level before the AE (Section 5.9.3.4). In the case of a serious discrepancy between the prescribed dose and the dose received, additional actions may be taken to modify data entries.

#### 5.9.3.4. Last Dose Level Prior to an Adverse Event

The last dose level prior to an AE is derived as the last non-zero dose (from EX domain) prior to the day an AE occurred. The reason to use "prior to the day" which excludes the day on which an AE occurred is that daily dose is divided into morning and evening doses and no dose administration time is collected on eCRF, making the last dose prior to an AE difficult to verify if "on the same day" dose levels are also included in the derivation.

It is noted that the data collected through the EX domain is treated as actual doses (rather than the prescribed dose schedule, as is the case of deriving compliance, defined earlier). This approach is used throughout when dose-response analyses (for both safety and efficacy) are carried out.

#### 5.9.4. Blood Transfusion Independence at Baseline

Transfusion independence at baseline is defined in 2 ways.

- 1. It is defined as receiving no transfusions (of red blood cell products) in the 8 weeks before Day 1.
- 2. It is defined as receiving no transfusions (of red blood cell products) in the 12 weeks before Day 1.

#### 5.9.5. Blood Transfusion Independence at Post-Baseline

Transfusion independence during post-baseline period is defined in 2 ways.

- 1. It is defined as receiving no transfusions (of red blood cell products) during the final 8 weeks of a subject's participation before the data cutoff date.
- 2. It is defined as receiving no transfusions (of red blood cell products) during the final 12 weeks of a subject's participation before the data cutoff date.

#### 5.9.6. Derivation of Per-protocol Population

The following process will be followed in deriving the PP population.

- Analysis programming team will generate a study drug compliance listing (by Week 24) and pass it to the clinical team.
- Based on study drug compliance and protocol deviation information from the clinical monitoring database, the clinical team will generate a PP population file indicating the membership of subjects to this population, and pass this file to the analysis programming team.
- Analysis programming team will use the PP population file to set the population indicator in analysis datasets for analysis.

In addition, the clinical team will also generate a source document containing all protocol deviations collected through the clinical monitoring process and pass it to the analysis programming team for generation of the protocol deviation listing.

# 6. BASELINE, EXPOSURE, AND DISPOSITION VARIABLES AND ANALYSES

# **6.1.** Baseline and Demographics

Descriptive summaries for demographic and baseline characteristics will include, but not limited to, age, age group ( $\leq$  65 vs > 65), sex, race, ethnicity, weight, height, ECOG performance status, transfusion history status, history of usage of any and all other drugs used to treat MF, and spleen palpation length. A data listing will be provided.

## **6.2.** Disposition and Enrollment

The number and percentage of subjects enrolled, completed, and withdrawn from the study with a primary reason of withdrawal will be summarized for the safety population. Per study design, disposition is applicable to the following 3 contexts: End of Treatment Phase or Early Termination, End of Extension Phase or Early Termination, and End of Study. Summaries will be provided for each of these 3 contexts and support listing will also be provided.

In addition, a listing for screen failures will be provided and will include information regarding demographics and eligibility status.

#### **6.3.** Protocol Deviations

Protocol deviations captured will be listed in subject data listings.

## 6.4. Exposure

For subjects in the safety population, descriptive statistics will be provided for duration of treatment (defined as days or weeks between first dose and last dose inclusive disregard dose interruptions in between); total patient years of exposure; total dose (mg); average daily dose (mg), which is defined as the total dose divided by duration of treatment; last titrated dose level (mg/day); and last average daily dose. Average daily dose (mg) will also be summarized by the major study time points (ie, during Weeks 1, 4, 8, 12, 16, 20, and 24). A data listing will be provided.

# **6.5.** Study Medication Compliance

Overall compliance (%) will be summarized and a data listing will be provided.

# 6.6. Medical History

Medical history will be summarized. Summaries will include the number and percentage of subjects with significant medical history for each body system/organ class listed on the CRF page.

#### 6.7. Concomitant Medication

Concomitant medications will be summarized by WHO drug class and WHO drug term. In the data listing, each record will be flagged as whether or not the medication is of prior, concomitant, or both prior and concomitant usage.

Prior medication information will also be reviewed by the clinical monitor to identify anti-cancer medication received by subjects prior to enrollment into the study. Prior anti-cancer medication data will be summarized as well as listed.

## **6.8.** Blood Transfusion Dependency

The proportion of subjects who were blood-transfusion dependent at baseline and at post-baseline will be summarized by baseline platelet count group (50-75 GI/L vs > 75 GI/L). A shift summary including the number and percentage of subjects who changed transfusion status was also produced by baseline platelet count group. In addition, the total units and average monthly units of transfusions will also be summarized by baseline platelet count group.

#### 7. EFFICACY ANALYSES

# 7.1. Primary Efficacy Endpoints

For the co-primary endpoints (correlation of percent change from baseline in spleen volume at Week 24 versus final titrated dose, and correlation of percent change from baseline in total symptom score at Week 24 versus final titrated dose), the following t-test will be used generate the p-values:

$$T = r \times \sqrt{\frac{n-2}{1-r^2}} \sim t_{n-2} \mid H_0$$

where r is the product-moment (Pearson) correlation coefficient, n is the sample size of paired observations, and  $\sim t_{n-2} \mid H_0$  means the test statistic will follow a t-distribution with n-2 degrees of freedom under the null hypothesis.

In addition, correlation estimate and the corresponding approximate 95% confidence intervals will be calculated by using the Fisher's *r*-to-*z* transformation. The following SAS codes will be used to generate the all these statistics:

```
ODS OUTPUT FisherPearsonCorr=correst PearsonCorr=pval;
PROC CORR FISHER PEARSON;
    VAR X Y;
RUN; ***CORREST has point estimate and CI from Fisher z-transformation, and
PVAL has p-value and the raw Pearson correlation coefficient ***;
```

The analysis will be generated for the ITT population. The same analysis will be repeated by using The PP population as a sensitivity analysis (Sensitivity Analysis 1).

An additional sensitivity analysis may be generated in dealing with missing data by using multiple imputation procedures (Sensitivity Analysis 2).

# 7.2. Secondary Endpoint(s) and Analyses

For the following secondary endpoints, descriptive summaries will be provided for overall as well as for the final titrated dose group:

- Percent change from baseline in spleen volume at Week 24.
- Percent change from baseline in total symptom score at Week 24.
- Proportion of subjects with ≥ 35% reduction from baseline in spleen volume at Week 24.
- Proportion of subjects with ≥ 10% reduction from baseline in spleen volume at Week 24.

- Proportion of subjects with  $\geq$  50% improvement from baseline in total symptom score at Week 24.
- Change and percentage change from baseline in spleen length as measured by palpation at each visit where the parameter is assessed.

Supporting data listings will also be provided.



#### 8. SAFETY ANALYSES

#### 8.1. Adverse Events

The following summaries will be produced for AEs for the overall subject group:

#### **High Level Summary**

- Number (%) of subjects reporting any TEAEs
- Number (%) of subjects reporting any DLT
- Number (%) of subjects reporting any treatment-related AEs
- Number (%) of subjects reporting any SAEs
- Number (%) of subjects reporting any Grade 3 or 4 AEs
- Number (%) of subjects who discontinued study drug because of AEs
- Number (%) of subjects with study drug dose reductions because of AEs
- Number (%) of subjects who died

#### By MedDRA Term:

- Number (%) of subjects reporting TEAEs by organ class and preferred term
- Number (%) of subjects reporting Grade 3 or 4 TEAEs by organ class and preferred term
- Number (%) of subjects reporting treatment-related AEs by organ class and preferred term
- Number (%) of subjects reporting treatment-emergent SAEs by organ class and preferred term
- Number (%) of subjects reporting treatment-emergent non-serious AEs by organ class and preferred term

In addition, a listing of DLTs will be provided.

These TEAEs occurring in 2 or more subjects in the safety population will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) preferred term for all causalities as well as for treatment-related causalities.

Proportion of subjects with new onset of Grade 4 thrombocytopenia events based on laboratory data and as measured by CTCAE grades will be summarized. The hazard function of time to onset of Grade 4 thrombocytopenia will be estimated using life table method.

Proportion of subjects with new onset of Grade 2 or higher hemorrhage based on preferred terms included in the Standardized MedDRA Query (SMQ) for "Haemorrhage terms (excluding laboratory terms) (SMQ)" and as measured by CTCAE grades will be summarized. The hazard functions of time to onset will be estimated using life table method.

Proportion of subjects with new onset of Grade 4 anemia based on laboratory data and as measured by CTCAE grades will be summarized. The hazard functions of time to onset will be estimated using life table method.

For the above 3 types of AEs, additional analyses using summary tables as well as data listings may be provided taking into account the blood transfusion status at baseline and post-baseline blood transfusion history.

Selected maximal severity AE summary tables will also be generated by the dose level the subject received.

## 8.2. Laboratory Values

Clinical laboratory tests including hematology, serum chemistry, coagulation, and urinalysis will be performed for each subject during the study in accordance with the Schedule of Observations (see Table 3). If specific safety issues arise, additional, unscheduled laboratory tests/analyses may be performed at the discretion of the investigator.

All test results and associated normal ranges from central laboratories will be reported in Standard International units (SI unit). All tests with numeric values will have a unique unit per test. Any laboratory results and associated normal ranges from local laboratories will be converted to SI units. When there are multiple laboratory values for a subject's particular test at a given visit, the last non-missing value will be used in the by-visit tabulations and summaries described below.

Numeric laboratory values will be summarized descriptively, and non-numeric test values will be tabulated by study visit using data collected from scheduled visits.

For those tests with available normal ranges, the number and percentage of subjects with the laboratory values being low, normal, or high will be calculated for each test. A shift summary will be produced, which presents the change from baseline as shown in Table 5.

Table 5:

| | | • | 1.1 | • | |
|---|---|---|---|---|---|
| | At a Post-baseline Visit | | | | |
| At Baseline | Missing | Low-Only | Normal | High-Only | Both Low and High |
| 3.4. | NI (0/) | NI (0/) | NI (0/) | NI (0/) | NI (0/) |

Missing N (%) Low N (%) N (%) Normal N (%) N (%) N (%) N (%) N (%) High N (%) N (%) N (%) N (%) N (%) Total N (%) N (%) N (%) N (%) N (100%)

**Example Shift Summary for Applicable Laboratory Assessments** 

Laboratory test values outside the normal range will be assessed for severity based on severity CTCAE grade or CTCAE grade criteria (where clinical intervention is required for CTCAE grading). Shift tables relative to baseline will be generated using all available data from scheduled and unscheduled visits.

#### 8.3. Vital Signs

Descriptive statistics for measurements, as well as change from baseline values, will be provided for vital signs (blood pressure, heart rate, respiratory rate, and body temperature) at each assessment time. Subjects exhibiting clinically notable vital sign abnormalities will be listed.

A value will be considered an "alert" value if it is outside the established range and shows a change from baseline greater than 25%, according to the high and/or low threshold values listed in Table 6.

High and Low Threshold Values for Alert Vital Sign Observations Table 6:

| Hg < 85 mm Hg |
|---------------------|
| Hg < 50 mm Hg |
| oute < 8 per minute |
| n < 45 bpm |

Alert vital sign data will also be listed.

#### **8.4. Electrocardiograms**

Electrocardiogram data collected at the screening visit will be listed. If additional data are collected, they will be listed and may be summarized as appropriate.

# 9. <u>CLINICAL PHARMACOLOGY</u>/



# 9.2. Subject Demographic, Clinical Laboratory, and Disease-Related Variables

Subject demographic assessments (age, weight, body mass index, sex, and race), disease-related evaluations (baseline platelet count, tumor type), and clinical laboratory measurements (creatinine clearance, ALB, total bilirubin, alkaline phosphatase, alanine aminotransferase, AST) may be explored as time independent predictors of variability.

#### 9.3. Concomitant Medication

CYP3A4 inhibitors and inducers may be may be tested as time dependent variables of variability if more than 15% of patients will take them as concomitant medications.





# 9.5. Pharmacokinetic-Pharmacodynamic Data Analysis

The relationship between PK model predicted concentrations/parameters and pharmacologic, safety, and efficacy read-outs are planned. A longitudinal analysis of platelets (absolute values or change from pre-dose) using predicted PK and baseline platelet values as covariates will be performed to assess platelet change over time. The population PK model will be used to derive estimates of individual steady-state exposure measures for PK-PD analysis.

## 9.6. Output

A population PK report will be prepared in accordance with guidance of both US and EU regulatory authorities.

## 10. LIST OF PLANNED TABLES, LISTINGS, AND FIGURES

#### **10.1.** Tables

| Table Number | Title | Population |
|---|---|---|
| Baseline and Demographic Characteristics | | |
| 14.1.1 | Summary of Subject Enrollment and Exit Status | Safety |
| 14.1.2 | Summary of Demographics | Safety |
| 14.1.3 | Summary of Baseline Characteristics | Safety |
| 14.1.4 | Summary of Medical History by MedDRA System Organ Class and Preferred Term | Safety |
| 14.1.5.1 | Summary of Prior Medications | Safety |
| 14.1.5.2 | Summary of Concomitant Medications | Safety |
| 14.1.5.3 | Summary of Prior Anti-Cancer Treatment | Safety |
| 14.1.6.1 | Summary of Change in Status of Blood Component Transfusion Dependency by Baseline Platelet Count Group | Safety |
| 14.1.6.2 | Summary of Blood Component Transfusions by Baseline Platelet Count<br>Group | Safety |
| <b>Efficacy</b> | | |
| 14.2.1.1 | Summary of Correlations of Final Titrated Dose vs. Percent Change | ITT |
| | from Baseline in Spleen Volume at Week 24 and vs. Percent Change | |
| | in Total Symptom Score at Week 24 | |

| Table Number | Title | Population |
|---|---|---|
| 14.2.1.2 | Summary of Correlations of Final Titrated Dose vs. Percent Change from Baseline in Spleen Volume at Week 24 and vs. Percent Change | Per-Protocol |
| 14.2.1.3 | in Total Symptom Score at Week 24: Sensitivity Analysis 1 Summary of Correlations of Final Titrated Dose vs. Percent Change from Baseline in Spleen Volume at Week 24 and vs. Percent Change in Total Symptom Score at Week 24: Sensitivity Analysis 2 | ITT |
| 14.2.2.1 | Summary of Spleen Volume Data by Study Week and Final Titrated Dose Group | ITT |
| 14.2.2.2 | Summary of Proportion of Subjects with >= 35% Reduction from Baseline in Spleen Volume at Week 24 by Final Titrated Dose Group | ITT |
| 14.2.2.3 | Summary of Proportion of Subjects with >= 10% Reduction from Baseline in Spleen Volume at Week 24 by Final Titrated Dose Group | ITT |
| 14.2.3.1 | Summary of Total Symptom Score Data by Study Week and Final Titrated Dose Group | ITT |
| 14.2.3.2 | Summary of Proportion of Subjects with >= 50% Reduction from Baseline in Total Symptom Score by Study Week and Final Titrated Dose Group | ITT |
| 14.2.4.1 | Summary of Spleen Palpation Length Data by Study Week and Final Titrated Dose Group | ITT |
| 14.2.4.2 | Summary of Proportion of Subjects with >= 50% Reduction from Baseline in Spleen Palpation Length by Study Week and Final Titrated Dose Group | ITT |
| 14.2.4.3 | Summary of Proportion of Subjects with >= 20% Reduction from Baseline in Spleen Palpation Length by Study Week and Final Titrated Dose Group | ITT |
| Safety: Exposur<br>14.3.1.1 | Summary of Exposure and Duration of Exposure to Study Medication Through Week 24 | Safety |
| 14.3.1.2 | Summary of Exposure to Ruxolitinib Through Week 4 | Safety |
| 14.3.1.3 | Summary of Average Daily Dose of Ruxolitinib by Study Week | Safety |
| Safety: Adverse | | |
| 14.3.2.1 | Overall Summary of Treatment-Emergent Adverse Events by Dose<br>Level Ever Received | Safety |
| 14.3.2.2.1 | Summary of Subjects Reporting Treatment-Emergent Adverse<br>Events (All Causalities) by MedDRA System Organ Class, Preferred<br>Term, and Maximum Severity | Safety |
| Table Number | Title | Population |
|---|---|---|
| 14.3.2.2.2 | Summary of Subjects Reporting Treatment-Emergent Adverse<br>Events (All Causalities) by MedDRA System Organ Class, Preferred<br>Term, and Dose Level Ever Received | Safety |
| 14.3.2.3.1 | Summary of Subjects Reporting Treatment-Emergent Adverse<br>Events (All Causalities) by MedDRA Preferred Term (Sorted by<br>Decreasing Frequency) and Maximal Severity | Safety |
| 14.3.2.3.2 | Summary of Subjects Reporting Treatment-Emergent Adverse<br>Events (All Causalities) by MedDRA Preferred Term (Sorted by<br>Decreasing Frequency) and Dose Level Ever Received | Safety |
| 14.3.2.3.3 | Summary of Subjects Reporting Treatment-Emergent Hemorrhage<br>Adverse Events (All Causalities) by MedDRA Preferred Term and<br>Dose Level Ever Received | Safety |
| 14.3.2.3.4 | Summary of Subjects Reporting Treatment-Emergent Hemorrhage<br>Adverse Events (All Causalities) of Grade 3 or Higher by MedDRA<br>Preferred Term and Dose Level Ever Received | Safety |
| 14.3.2.4.1 | Summary of Subjects Reporting Treatment-Emergent Treatment-Related Adverse Events (All Causalities) by MedDRA System Organ Class, Preferred Term, and Maximum Severity | Safety |
| 14.3.2.4.2 | Summary of Subjects Reporting Treatment-Emergent Treatment-Related Adverse Events (All Causalities) by MedDRA System Organ Class, Preferred Term, and Dose Level Ever Received | Safety |
| 14.3.2.5.1 | Summary of Subjects Reporting Treatment-Emergent Serious<br>Adverse Events (All Causalities) by MedDRA System Organ Class,<br>Preferred Term, and Dose Level Ever Received | Safety |
| 14.3.2.6 | Summary of Subjects Reporting Treatment-Emergent Adverse<br>Events (All Causalities) Leading to Study Medication Decrease or<br>Interruption by MedDRA System Organ Class, Preferred Term, and<br>Dose Level Ever Received | Safety |
| 14.3.2.7 | Summary of Subjects Reporting Treatment-Emergent Adverse<br>Events (All Causalities) Leading to Study Discontinuation by<br>MedDRA System Organ Class, Preferred Term, and Dose Level<br>Ever Received | Safety |
| 14.3.2.8 | Summary of Subjects Reporting Treatment-Emergent Adverse<br>Events (All Causalities) Leading to On-Study Death by MedDRA<br>System Organ Class, Preferred Term, and Dose Level Ever<br>Received | Safety |
| Safety: Laborat | ory Data | |
| 14.3.3.1.1 | Summary of Laboratory Values – Hematology | Safety |
| 14.3.3.1.2 | Shift Summary of Laboratory Values in Normal Ranges -<br>Hematology | Safety |
| 14.3.3.2.1 | Summary of Laboratory Values – Serum Chemistry | Safety |
| 14.3.3.2.2 | Shift Summary of Laboratory Values in Normal Ranges – Serum Chemistry | Safety |
| 14.3.3.3.1 | Summary of Laboratory Values – Coagulation | Safety |
| 14.3.3.3.2 | Shift Summary of Laboratory Values in Normal Ranges – Coagulation | Safety |
| 14.3.3.4.1 | Summary of Laboratory Values – Urinalysis | Safety |
| 14.3.3.4.2 | Shift Summary of Laboratory Values in Normal Ranges – Urinalysis | Safety |
| 14.3.3.5.1 | Shift Summary of Laboratory Values in CTC Grade - To the Worst Abnormal Value (Tests with One Directional CTC Grade) | Safety |

| Table Number | Title | Population |
|---|---|---|
| 14.3.3.5.2 | Shift Summary of Laboratory Values in CTC Grade - To the Worst | Safety |
| | Abnormal Value (Tests with Two Directional CTC Grade) | - |
| 14.3.3.6.1 | Summary of Subjects with Treatment Emergent Thrombocytopenia | Safety |
| | of Grade 4 as Derived From Laboratory Data by Dose Level Ever | - |
| | Received | |
| 14.3.3.6.2 | Summary of Subjects with Treatment Emergent Anemia of Grade 4 | Safety |
| | as Derived From Laboratory Data by Dose Level Ever Received | - |
| Safety: Vital Sig | <u>ins</u> | |
| 14.3.4.1 | Summary of Systolic Blood Pressure | Safety |
| 14.3.4.2 | Summary of Diastolic Blood Pressure | Safety |
| 14.3.4.3 | Summary of Heart Rate | Safety |
| 14.3.4.4 | Summary of Respiratory Rate | Safety |
| 14.3.4.5 | Summary of Body Temperature | Safety |

10.2. Figures

| 10.4. | rigures | |
|---|---|---|
| Figure<br>Number | Title | Population |
| 14.2.1.1.1 | Scatter Plot of Percent Change from Baseline in Spleen Volume at Week 24 vs. Final Titrated Dose Level | ITT |
| 14.2.1.1.2 | Scatter Plot of Percent Change from Baseline in Spleen Volume vs. Percent Change in Total Symptom Score at Week 24 | ITT |
| 14.2.1.2.1 | Mean (95%) Percent Change from Baseline in Spleen Volume at Week 24 | ITT |
| 14.2.1.2.2 | Median Percent Change from Baseline in Spleen Volume at Week 24 by Final Titrated Dose Group | ITT |
| 14.2.1.3.1 | Bar Plot of Percent of Subjects with >= 35% Reduction from Baseline in Spleen Volume at Week 24 by Final Titrated Dose Group | ITT |
| 14.2.1.3.2 | Bar Plot of Percent of Subjects with >= 10% Reduction from Baseline in Spleen Volume at Week 24 by Final Titrated Dose Group | ITT |
| 14.2.2.1.1 | Scatter Plot of Percent Change from Baseline in Total Symptom<br>Score at Week 24 vs. Final Titrated Dose Level | ITT |
| 14.2.2.2.1 | Mean (95%) Percent Change from Baseline in Total Symptom Score at Week 24 by Final Titrated Dose Group | ITT |
| 14.2.2.2.2 | Median Percent Change from Baseline in Total Symptom Score at Week 24 by Final Titrated Dose Group | ITT |
| 14.2.2.3.1 | Bar Plot of Percent of Subjects with >= 50% Reduction from Baseline in Total Symptom Score at Week 24 by Final Titrated Dose Group | ITT |
| 14.2.3.1.1 | Scatter Plot of Percent Change from Baseline in Spleen Palpation<br>Length at Week 24 vs. Final Titrated Dose Level | ITT |
| 14.2.3.2.1 | Mean (95%) Percent Change from Baseline in Spleen Palpation<br>Length at Week 24 by Final Titrated Dose Group | ITT |
| 14.2.3.2.2 | Median Percent Change from Baseline in Spleen Palpation Length at Week 24 by Final Titrated Dose Group | ITT |

| Figure | | |
|---|---|---|
| Number | Title | Population |
| 14.2.3.3.1 | Bar Plot of Percent of Subjects with >= 50% Reduction from | ITT |
| | Baseline in Spleen Palpation Length at Week 24 by Final Titrated | |
| | Dose Group | |
| 14.2.3.3.2 | Bar Plot of Percent of Subjects with >= 20% Reduction from | ITT |
| | Baseline in Spleen Palpation Length at Week 24 by Final Titrated | |
| | Dose Group | |
| 14.2.3.3.3 | Bar Plot of Percent of Subjects with >= 50% Reduction from | ITT |
| | Baseline in Spleen Palpation Length by Study Week | |
| 14.2.3.3.4 | Bar Plot of Percent of Subjects with >= 20% Reduction from | ITT |
| | Baseline in Spleen Palpation Length at Week 24 by Study Week | |
| 14.3.1.1.1 | Subject Laboratory Value over Time: Hemoglobin (G/L) | Safety |
| 14.3.1.1.2 | Mean (95% CI) Laboratory Value Over Time: Hemoglobin (G/L) | Safety |
| 14.3.1.2.1 | Subject Laboratory Value over Time: Platelet (GI/L) | Safety |
| 14.3.1.2.2 | Mean (95% CI) Laboratory Value Over Time: Platelet (GI/L) | Safety |
| 14.3.1.3.1 | Subject Laboratory Value over Time: WBC (GI/L) | Safety |
| 14.3.1.3.2 | Mean (95% CI) Laboratory Value Over Time: WBC (GI/L) | Safety |
| 14.3.1.4.1 | Subject Laboratory Value over Time: Neutrophil (GI/L) | Safety |
| 14.3.1.4.2 | Mean (95% CI) Laboratory Value Over Time: Neutrophil (GI/L) | Safety |

10.3. Listings

| Listing | | |
|---|---|---|
| Number | Title | Population |
| 16.2.1.1 | Subject Enrollment and Exit Status | Safety |
| 16.2.1.2 | Screening Failure Subjects | Safety |
| 16.2.2 | Protocol Deviations/Violations | Safety |
| 16.2.3 | Data Excluded from Efficacy, and/or Safety Analyses | Safety |
| 16.2.4.1 | Demographic and Baseline Characteristics | Safety |
| 16.2.4.2.1 | Medical History | Safety |
| 16.2.4.2.2 | Baseline Disease Stage | Safety |
| 16.2.4.3 | Prior and Concomitant Drug Treatments | Safety |
| 16.2.4.4 | Prior Myelofibrosis Therapy | Safety |
| 16.2.4.5 | Prior Anti-Cancer Treatment | Safety |
| 16.2.6.1 | Derived Efficacy Variables – Part I | ITT |
| 16.2.6.2 | Derived Efficacy Variables – Part II | ITT |
| 16.2.7.1.1 | Study Drug Activities and Dosing Compliance | Safety |
| 16.2.7.2.1 | Adverse Events | Safety |
| 16.2.7.2.2 | Serious Adverse Events | Safety |
| 16.2.7.2.3 | Adverse Event Leading to Study Drug Decrease, Interruption, and | Safety |
| | Discontinuation | |
| 16.2.7.2.4 | Adverse Events of Hemorrhage as Identified by SMQ | Safety |
| 16.2.7.2.5 | Adverse Events Leading to Discontinuation from the Study | Safety |
| 16.2.7.2.6 | Adverse Events Leading to On-Study Death | Safety |
| 16.2.8.1.1 | Clinical Laboratory Values | Safety |
| 16.2.8.1.2 | Abnormal Clinical Laboratory Values | Safety |
| 16.2.8.1.3 | Selected Hematology Laboratory Data | Safety |
| 16.2.8.1.4 | Selected Hematology Laboratory Data for Subjects with Grade 4<br>Thrombocytopenia or Grade 4 Anemia | Safety |

| Listing | | |
|------------|--------------------------------------|------------|
| Number | Title | Population |
| 16.2.8.2.1 | Vital Signs | Safety |
| 16.2.8.2.2 | Abnormal Vital Sign Values | Safety |
| 16.2.8.2.3 | Alert Vital Sign Values | |
| 16.2.8.3.1 | 12-Lead ECG Values | Safety |
| 16.2.8.3.2 | Abnormal 12-Lead ECG Values | Safety |
| 16.2.8.4 | Physical Examinations | Safety |
| 16.2.8.5 | 6.2.8.5 Blood Component Transfusions | |
| 16.2.8.6 | Serum Pregnancy Test | Safety |

#### 11. REFERENCES

INCB18424-2581 Protocol Amendment 1.

- US Department of Health and Human Services, "Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03" 2010.
- http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE 4.03 2010-06-14 QuickReference 5x7.pdf
- CTEP, National Cancer Institute Drug Branch, "CTEP Guidance: CTCAE v4.0 Grading Scales with Numeric Component" 2010.
  - http://evs.nci.nih.gov/ftp1/CTCAE/Documentation/CTEP\_Guidance\_Quant-Grade\_2010-05-17.doc
- US FDA, "Guidance for Industry: Clinical Trial Endpoints for the Approval of Cancer Drugs and Biologics" 2007.
- SAS/STAT User Guides, Version 9.
- Cohen J: Statistical Power Analysis for the Behavioral Sciences. Second Edition. Hillsdale, NJ, 1988.

### 12. APPENDICES

# APPENDIX A. MEDDRA PREFERRED TERMS INCLUDED IN THE SMQ TO IDENTIFY HEMORRHAGE ADVERSE EVENTS

| Name | Code | Level | Scope | Cate-<br>gory | Weight | Status | Add.<br>Ver. | Last<br>Mod.<br>Ver. |
|---|---|---|---|---|---|---|---|---|
| Abdominal wall haematoma | 10067383 | PT | Narrow | A | 0 | Active | 10.1 | 12 |
| Abdominal wall haemorrhage | 10067788 | PT | Narrow | Α | 0 | Active | 11 | 12 |
| Abnormal withdrawal bleeding | 10069195 | PT | Narrow | Α | 0 | Active | 12 | 12 |
| Acute haemorrhagic | | | | | | | | |
| leukoencephalitis | 10058994 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Adrenal haematoma | 10059194 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Adrenal haemorrhage | 10001361 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Anal haemorrhage | 10049555 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Anal ulcer haemorrhage | 10063896 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Anastomotic haemorrhage | 10056346 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Anastomotic ulcer haemorrhage | 10002244 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Aneurysm ruptured | 10048380 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Anorectal varices haemorrhage | 10068925 | PT | Narrow | A | 0 | Active | 12 | 12 |
| Antepartum haemorrhage | 10002667 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Aortic aneurysm rupture | 10002886 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Aortic dissection rupture | 10068119 | PT | Narrow | A | 0 | Active | 11 | 12 |
| Aortic intramural haematoma | 10067975 | PT | Narrow | Α | 0 | Active | 11 | 12 |
| Aortic rupture | 10060874 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Application site bleeding | 10048938 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Application site haematoma | 10068317 | PT | Narrow | A | 0 | Active | 11.1 | 12 |
| Arterial haemorrhage | 10060964 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Arteriovenous fistula site haematoma | 10055150 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Arteriovenous fistula site haemorrhage | 10055123 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Arteriovenous graft site haematoma | 10055152 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Arteriovenous graft site haemorrhage | 10055126 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Astringent therapy | 10067372 | PT | Narrow | A | 0 | Active | 10.1 | 12 |
| Atrial rupture | 10048761 | PT | Narrow | A | 0 | Active | 13 | 13 |
| Auricular haematoma | 10003797 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Basal ganglia haemorrhage | 10067057 | PT | Narrow | A | 0 | Active | 10 | 12 |
| Bladder tamponade | 10062656 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Bleeding peripartum | 10048607 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Bleeding varicose vein | 10005144 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Blood blister | 10005372 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Blood urine | 10005863 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Blood urine present | 10018870 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Bloody discharge | 10057687 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Bloody peritoneal effluent | 10067442 | PT | Narrow | A | 0 | Active | 10.1 | 12 |
| Brain stem haemorrhage | 10006145 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Breast haematoma | 10064753 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Breast haemorrhage | 10006254 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Broad ligament haematoma | 10006375 | PT | Narrow | A | 0 | Active | 9 | 12 |

| Nama | Codo | Lavel | Saana | Cate- | Weight | Status | Add.<br>Ver. | Last<br>Mod.<br>Ver. |
|---|---|---|---|---|---|---|---|---|
| Name Bronchial haemorrhage | <b>Code</b> 10065739 | Level<br>PT | Scope<br>Narrow | gory<br>A | 0 | Active | 9 | 12 |
| Carotid aneurysm rupture | 10063739 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Catheter site haematoma | 10051528 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Catheter site haemorrhage | 10053002 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Cephalhaematoma | 10031099 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Cerebellar haematoma | 10061038 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Cerebellar haemorrhage | 10001038 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Cerebral aneurysm ruptured syphilitic | 10008030 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Cerebral arteriovenous malformation haemorrhagic | 10008086 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Cerebral haematoma | 10053942 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Cerebral haemorrhage | 10008111 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Cerebral haemorrhage foetal | 10050157 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Cerebral haemorrhage neonatal | 10008112 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Cerebral haemorrhage traumatic | 10008113 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Cerebral microhaemorrhage | 10067277 | PT | Narrow | A | 0 | Active | 10 | 12.1 |
| Cervix haematoma uterine | 10050020 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Cervix haemorrhage uterine | 10050022 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Choroidal haematoma | 10068642 | PT | Narrow | A | 0 | Active | 11.1 | 12 |
| Choroidal haemorrhage | 10008786 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Chronic gastrointestinal bleeding | 10050399 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Ciliary body haemorrhage | 10057417 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Coital bleeding | 10065019 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Colonic haematoma | 10009996 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Conjunctival haemorrhage | 10010719 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Contusion | 10050584 | PT | Narrow | A | 0 | Active | 13 | 13 |
| Corneal bleeding | 10051558 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Cullen's sign | 10059029 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Cystitis haemorrhagic | 10011793 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Diarrhoea haemorrhagic | 10012741 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Disseminated intravascular coagulation | 10013442 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Diverticulitis intestinal haemorrhagic | 10013541 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Diverticulum intestinal haemorrhagic | 10013560 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Duodenal ulcer haemorrhage | 10013839 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Duodenitis haemorrhagic | 10013865 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Dysfunctional uterine bleeding | 10013908 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Ear haemorrhage | 10014009 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Ecchymosis | 10014080 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Encephalitis haemorrhagic | 10014589 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Enterocolitis haemorrhagic | 10014896 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Epistaxis | 10015090 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Exsanguination | 10015719 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Extradural haematoma | 10015769 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Extravasation blood | 10015867 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Eye haemorrhage | 10015926 | PT | Narrow | A | 0 | Active | 9 | 12 |

| Name | Code | Level | Scope | Cate-<br>gory | Weight | Status | Add.<br>Ver. | Last<br>Mod.<br>Ver. |
|---|---|---|---|---|---|---|---|---|
| Eyelid bleeding | 10053196 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Foetal-maternal haemorrhage | 10035170 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Gastric haemorrhage | 10017788 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Gastric ulcer haemorrhage | 10017826 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Gastric ulcer haemorrhage, | 10017020 | | 11411011 | | Ů | 1100170 | | - 12 |
| obstructive | 10017829 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Gastric ulcer perforation | 10017835 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Gastric varices haemorrhage | 10057572 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Gastritis alcoholic haemorrhagic | 10017857 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Gastritis haemorrhagic | 10017866 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Gastroduodenal haemorrhage | 10053768 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Gastroduodenitis haemorrhagic | 10048712 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Gastrointestinal angiodysplasia haemorrhagic | 10017929 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Gastrointestinal haemorrhage | 10017955 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Gastrointestinal ulcer haemorrhage | 10056743 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Genital haemorrhage | 10061178 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Gingival bleeding | 10018276 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Graft haemorrhage | 10063577 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Haemarthrosis | 10018829 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Haematemesis | 10018830 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Haematochezia | 10018836 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Haematoma | 10018852 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Haematoma evacuation | 10060733 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haematoma infection | 10051564 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haematomyelia | 10066960 | PT | Narrow | A | 0 | Active | 10 | 12 |
| Haematosalpinx | 10050468 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haematospermia | 10018866 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haematotympanum | 10063013 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haematuria | 10018867 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haematuria traumatic | 10018871 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemobilia | 10058947 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Haemophilic arthropathy | 10065057 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Haemoptysis | 10018964 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Haemorrhage | 10055798 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Haemorrhage coronary artery | 10055803 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Haemorrhage foetal | 10061191 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Haemorrhage intracranial | 10018985 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Haemorrhage neonatal | 10061993 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhage subcutaneous | 10018999 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhage subepidermal | 10019001 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhage urinary tract | 10055847 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhagic anaemia | 10052293 | PT | Narrow | A | 0 | Active | 9.1 | 12 |
| Haemorrhagic arteriovenous malformation | 10064595 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhagic ascites | 10059766 | PT | Narrow | A | 0 | Active | 9 | 12 |

| Name | Code | Level | Scope | Cate-<br>gory | Weight | Status | Add.<br>Ver. | Last<br>Mod.<br>Ver. |
|---|---|---|---|---|---|---|---|---|
| Haemorrhagic cerebral infarction | 10019005 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhagic diathesis | 10062713 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhagic disease of newborn | 10019008 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhagic disorder | 10019009 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhagic erosive gastritis | 10067786 | PT | Narrow | A | 0 | Active | 11 | 12 |
| Haemorrhagic hepatic cyst | 10067796 | PT | Narrow | A | 0 | Active | 11 | 12 |
| Haemorrhagic infarction | 10019013 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhagic ovarian cyst | 10060781 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhagic stroke | 10019016 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhagic transformation stroke | 10055677 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhagic tumour necrosis | 10054096 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhagic urticaria | 10059499 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemorrhoidal haemorrhage | 10054787 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Haemostasis | 10067439 | PT | Narrow | A | 0 | Active | 10.1 | 12 |
| Haemothorax | 10019027 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Henoch-Schonlein purpura | 10019617 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Hepatic haemangioma rupture | 10054885 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Hepatic haematoma | 10019676 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Hepatic haemorrhage | 10019677 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Hereditary haemorrhagic telangiectasia | 10019883 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Hyphaema | 10020923 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Implant site haematoma | 10063780 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Implant site haemorrhage | 10053995 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Incision site haematoma | 10059241 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Incision site haemorrhage | 10051100 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Increased tendency to bruise | 10021688 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Induced abortion haemorrhage | 10052844 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Infusion site haematoma | 10065463 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Infusion site haemorrhage | 10065464 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Injection site haematoma | 10022066 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Injection site haemorrhage | 10022067 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Intestinal haemorrhage | 10059175 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Intra-abdominal haematoma | 10056457 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Intra-abdominal haemorrhage | 10061249 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Intracerebral haematoma evacuation | 10062025 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Intracranial haematoma | 10059491 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Intracranial tumour haemorrhage | 10022775 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Intrapartum haemorrhage | 10067703 | PT | Narrow | A | 0 | Active | 10.1 | 12 |
| Intraventricular haemorrhage | 10022840 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Intraventricular haemorrhage | 10022041 | DT | NT. | | | , | | 10 |
| neonatal | 10022841 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Iris haemorrhage | 10057418 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Lacrimal haemorrhage | 10069930 | PT | Narrow | A | 0 | Active | 13 | 13 |
| Large intestinal haemorrhage | 10052534 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Large intestinal ulcer haemorrhage | 10061262 | PT | Narrow | A | 0 | Active | 9 | 12 |

| Name | Code | Level | Scope | Cate-<br>gory | Weight | Status | Add.<br>Ver. | Last<br>Mod.<br>Ver. |
|---|---|---|---|---|---|---|---|---|
| Laryngeal haemorrhage | 10065740 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Lip haematoma | 10066304 | PT | Narrow | A | 0 | Active | 9.1 | 12 |
| Lip haemorrhage | 10049297 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Lower gastrointestinal haemorrhage | 10050953 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Majocchi's purpura | 10052316 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Mallory-Weiss syndrome | 10026712 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Mediastinal haematoma | 10049941 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Mediastinal haemorrhage | 10056343 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Melaena | 10027141 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Melaena neonatal | 10049777 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Meningorrhagia | 10052593 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Menometrorrhagia | 10027295 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Menorrhagia | 10027313 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Metrorrhagia | 10027514 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Mouth haemorrhage | 10028024 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Mucosal haemorrhage | 10061298 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Muscle haemorrhage | 10028309 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Myocardial haemorrhage | 10028309 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Myocardial rupture | 10048649 | PT | Narrow | A | 0 | Active | 13 | 13 |
| Naevus haemorrhage | 10028004 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Nail bed bleeding | 10002933 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Nephritis haemorrhagic | 10048331 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Nipple exudate bloody | 10029132 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Ocular retrobulbar haemorrhage | 10029418 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Oesophageal haemorrhage | 10037371 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Oesophageal ulcer haemorrhage | 10030172 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Oesophageal varices haemorrhage | 10030202 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Oesophagitis haemorrhagic | 10030210 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Operative haemorrhage | 10030219 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Optic disc haemorrhage | 10030800 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Optic nerve sheath haemorrhage | 10030919 | PT | Narrow | | 0 | Active | 9 | 12 |
| Osteorrhagia | 10050941 | PT | Narrow | A<br>A | 0 | Active | 9 | 12 |
| Ovarian haematoma | 10031937 | PT | | A | 0 | Active | 9 | 12 |
| Ovarian haemorrhage | 10055265 | PT | Narrow<br>Narrow | | | | 9 | 12 |
| Pancreatic haemorrhage | 10063741 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Pancreatitis haemorrhagic | 10033623 | PT | | A | 0 | Active | 9 | 12 |
| - | 10053630 | | Narrow | A | 0 | Active | 9 | |
| Papillary muscle haemorrhage Paranasal sinus haematoma | | PT | Narrow | A | | Active | | 12 |
| | 10069702 | PT | Narrow | A | 0 | Active | 13 | 13 |
| Parathyroid haemorrhage | 10059051 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Parotid gland haemorrhage | 10051166 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Pelvic haematoma | 10054974 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Pelvic haematoma obstetric | 10034248 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Pelvic haemorrhage | 10063678 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Penile haemorrhage | 10034305 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Peptic ulcer haemorrhage | 10034344 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Pericardial haemorrhage | 10034476 | PT | Narrow | Α | 0 | Active | 9 | 12 |

| Name | Code | Level | Scono | Cate- | Weight | Status | Add.<br>Ver. | Last<br>Mod.<br>Ver. |
|---|---|---|---|---|---|---|---|---|
| Perineal haematoma | 10034520 | PT | Scope<br>Narrow | gory<br>A | 0 | Active | 9 | 12 |
| Periorbital haematoma | 10034520 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Perirenal haematoma | 10034344 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Peritoneal haematoma | 10049430 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Peritoneal haemorrhage | 10034666 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Petechiae | 10034000 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Pharyngeal haematoma | 10068121 | PT | Narrow | A | 0 | Active | 11 | 12 |
| Pharyngeal haemorrhage | 10034827 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Pituitary haemorrhage | 10034827 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Placenta praevia haemorrhage | 10049700 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Pleural haemorrhage | 10035121 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Polymenorrhagia | 10033001 | PT | Narrow | A | 0 | Active | 9 | 12 |
| | + | PT | | | 0 | | 9 | 12 |
| Post abortion haemorrhage | 10036246 | | Narrow | A | 0 | Active | 9 | |
| Post procedural haematoma | | PT | Narrow | A | - | Active | | 12 |
| Post procedural haematuria | 10066225 | PT | Narrow | A | 0 | Active | 9.1 | 12 |
| Post procedural haemorrhage | 10051077 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Postmenopausal haemorrhage | 10055870 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Postpartum haemorrhage | 10036417 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Premature separation of placenta | 10036608 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Proctitis haemorrhagic | 10036778 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Prostatic haemorrhage | 10036960 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Pulmonary alveolar haemorrhage | 10037313 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Pulmonary haematoma | 10054991 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Pulmonary haemorrhage | 10037394 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Puncture site haemorrhage | 10051101 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Purpura | 10037549 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Purpura neonatal | 10037557 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Purpura senile | 10037560 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Putamen haemorrhage | 10058940 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Rectal haemorrhage | 10038063 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Rectal ulcer haemorrhage | 10038081 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Renal cyst haemorrhage | 10059846 | PT | Narrow | A | 0 | Active | 9 | 13 |
| Renal haematoma | 10038459 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Renal haemorrhage | 10038460 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Respiratory tract haemorrhage | 10038727 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Respiratory tract haemorrhage neonatal | 10038728 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Retinal haemorrhage | 10038728 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Retinopathy haemorrhagic | 10058807 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Retroperitoneal haematoma | 10051447 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Retroperitoneal haematoma Retroperitoneal haemorrhage | 10038360 | PT | | A | 0 | | 9 | 12 |
| Retroperitoneal naemorrnage Retroplacental haematoma | 10038980 | PT | Narrow<br>Narrow | A | 0 | Active Active | 9 | 12 |
| • | 10034798 | PT | | | 0 | | 9 | 12 |
| Ruptured cerebral aneurysm Scleral haemorrhage | 1 | PT<br>PT | Narrow<br>Narrow | A | 0 | Active | 9 | 12 |
| Scieral naemorrnage Scrotal haematocoele | 10050508<br>10061517 | PT | | A | 0 | Active | 9 | 12 |
| | | | Narrow | A | | Active | | |
| Scrotal haematoma | 10039749 | PT | Narrow | A | 0 | Active | 9 | 12 |

| Nome | Code | Lovel | Saona | Cate- | Weight | Status | Add. | Last<br>Mod.<br>Ver. |
|---|---|---|---|---|---|---|---|---|
| Name Shock haemorrhagic | 10049771 | Level<br>PT | Scope<br>Narrow | gory<br>A | 0 | Status<br>Active | Ver. | 12 |
| Skin haemorrhage | 10049771 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Skin ulcer haemorrhage | 10004203 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Small intestinal haemorrhage | 10030377 | PT | Narrow | A | 0 | | 9 | 12 |
| Small intestinal naemorrnage Small intestinal ulcer haemorrhage | 10052535 | PT | Narrow | A | 0 | Active<br>Active | 9 | 12 |
| · · | 10061330 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Soft tissue haemorrhage | | | | | - | | 9 | |
| Spermatic cord haemorrhage | 10065742 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Spinal cord haemorrhage | 10048992 | PT | Narrow | A | 0 | Active | | 12 |
| Spinal epidural haemorrhage | 10049236 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Spinal haematoma | 10048464 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Splenic haematoma | 10041646 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Splenic haemorrhage | 10041647 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Splenic varices haemorrhage | 10068662 | PT | Narrow | A | 0 | Active | 11.1 | 12 |
| Splinter haemorrhages | 10041663 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Spontaneous haematoma | 10065304 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Stomatitis haemorrhagic | 10042132 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Subarachnoid haemorrhage | 10042316 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Subarachnoid haemorrhage neonatal | 10042317 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Subcutaneous haematoma | 10042345 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Subdural haematoma | 10042361 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Subdural haematoma evacuation | 10042363 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Subdural haemorrhage | 10042364 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Subdural haemorrhage neonatal | 10042365 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Subgaleal haematoma | 10069510 | PT | Narrow | A | 0 | Active | 12.1 | 12.1 |
| Testicular haemorrhage | 10051877 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Thalamus haemorrhage | 10058939 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Third stage postpartum haemorrhage | 10043449 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Thoracic haemorrhage | 10062744 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Thrombocytopenic purpura | 10043561 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Thrombotic thrombocytopenic | | | | | | | | |
| purpura | 10043648 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Thyroid haemorrhage | 10064224 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Tongue haematoma | 10043959 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Tongue haemorrhage | 10049870 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Tonsillar haemorrhage | 10057450 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Tooth socket haemorrhage | 10064946 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Tracheal haemorrhage | 10062543 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Traumatic haematoma | 10044522 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Traumatic haemorrhage | 10053476 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Traumatic intracranial haemorrhage | 10061387 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Tumour haemorrhage | 10049750 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Ulcer haemorrhage | 10061577 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Umbilical cord haemorrhage | 10064534 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Umbilical haematoma | 10068712 | PT | Narrow | A | 0 | Active | 11.1 | 12 |
| Umbilical haemorrhage | 10045455 | PT | Narrow | Α | 0 | Active | 9 | 12 |
| Upper gastrointestinal haemorrhage | 10046274 | PT | Narrow | A | 0 | Active | 9 | 12 |

| Name | Code | Level | Scope | Cate-<br>gory | Weight | Status | Add.<br>Ver. | Last<br>Mod.<br>Ver. |
|---|---|---|---|---|---|---|---|---|
| Ureteric haemorrhage | 10065743 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Urethral haemorrhage | 10049710 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Urinary bladder haemorrhage | 10046528 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Urogenital haemorrhage | 10050058 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Uterine haematoma | 10063875 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Uterine haemorrhage | 10046788 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Vaccination site haematoma | 10069472 | PT | Narrow | A | 0 | Active | 12.1 | 12.1 |
| Vaccination site haemorrhage | 10069475 | PT | Narrow | A | 0 | Active | 12.1 | 12.1 |
| Vaginal haematoma | 10046909 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Vaginal haemorrhage | 10046910 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Varicose vein ruptured | 10046999 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Vascular pseudoaneurysm ruptured | 10053949 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Vascular purpura | 10047097 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Vascular rupture | 10053649 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Venous haemorrhage | 10065441 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Ventricle rupture | 10047279 | PT | Narrow | A | 0 | Active | 13 | 13 |
| Vessel puncture site haematoma | 10065902 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Vessel puncture site haemorrhage | 10054092 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Vitreous haemorrhage | 10047655 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Vulval haematoma | 10047756 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Vulval haematoma evacuation | 10047757 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Vulval haemorrhage | 10063816 | PT | Narrow | A | 0 | Active | 9 | 12 |
| Wound haemorrhage | 10051373 | PT | Narrow | A | 0 | Active | 9 | 12 |

### APPENDIX B. SHELLS FOR POST-TEXT TABLES

Shells for post-text tables are presented starting from next page.

PROTOCOL: INCB 18424-258 
DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.1

Summary of Subject Enrollment and Exit Status (Population: Safety Evaluable Subjects)

| Variable | Ruxolitinib<br>(N=xxx) |
|---|---|
| <br>Number (%) of Subjects Completed Treatment Phase | xxx ( xx.x) |
| Number (%) of Subjects Entered Extension Phase | xxx ( xx.x) |
| Number (%) of Subjects Still on Study | xxx ( xx.x) |
| Number (%) of Subjects Discontinued During Treatment Phase | xxx ( xx.x) |
| Primary Reason of Discontinuation: Treatment Phase | |
| Death | xxx ( xx.x) |
| Adverse Event | xxx ( xx.x) |
| Consent Withdrawn | xxx ( xx.x) |
| Protocol Deviation | xxx ( xx.x) |
| Disease Progression | xxx ( xx.x) |
| Lost to Follow-up | xxx ( xx.x) |
| Non-Compliance with Study Medication | xxx ( xx.x) |
| Non-Compliance with Study Procedures | xxx ( xx.x) |
| Termination of the Clinical Trial by the Sponsor | xxx ( xx.x) |

PROGRAM\OUTPUT: T\_DISP.SAS\T\_TERM1.LST

DATE(TIME): DDMMMYY(HH:MM)

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.1

Summary of Subject Enrollment and Exit Status (Population: Safety Evaluable Subjects)

| ** 11 | Ruxolitinib |
|------------------------------------------------------------|-------------|
| Variable | (N=xxx) |
| Number (%) of Subjects Discontinued During Extension Phase | xxx ( xx.x) |
| Primary Reason of Discontinuation: Extension Phase | |
| Death | xxx ( xx.x) |
| Adverse Event | xxx ( xx.x) |
| Consent Withdrawn | xxx ( xx.x) |
| Protocol Deviation | xxx ( xx.x) |
| Disease Progression | xxx ( xx.x) |
| Lost to Follow-up | xxx ( xx.x) |
| Non-Compliance with Study Medication | xxx ( xx.x) |
| Non-Compliance with Study Procedures | xxx ( xx.x) |
| Termination of the Clinical Trial by the Sponsor | xxx ( xx.x) |
| Other | xxx ( xx.x) |

PROGRAM\OUTPUT: T DISP.SAS\T TERM1.LST

DATE(TIME): DDMMMYY(HH:MM)

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.1

Summary of Subject Enrollment and Exit Status (Population: Safety Evaluable Subjects)

| Variable | Ruxolitinib<br>(N=xxx) |
|---|---|
| Number (%) of Subjects Discontinued During the Study | xxx ( xx.x) |
| Primary Reason of Discontinuation: Extension Phase | |
| Death | xxx ( xx.x) |
| Adverse Event | xxx ( xx.x) |
| Consent Withdrawn | xxx ( xx.x) |
| Protocol Deviation | xxx ( xx.x) |
| Disease Progression | xxx ( xx.x) |
| Lost to Follow-up | xxx ( xx.x) |
| Non-Compliance with Study Medication | xxx ( xx.x) |
| Non-Compliance with Study Procedures | xxx ( xx.x) |
| Termination of the Clinical Trial by the Sponsor | xxx ( xx.x) |
| Other | xxx ( xx.x) |

PROGRAM\OUTPUT: T\_DISP.SAS\T\_TERM1.LST

DATE(TIME): DDMMMYY(HH:MM)

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.2

# Summary of Demographics (Population: Safety Evaluable Subjects)

| Ruxolitinib | |
|-------------------------------------|-------------|
| Variable | (N=xxx) |
| Age (yrs) | |
| n | XXX |
| Mean | XX.X |
| STD | X.XX |
| Min | XX.X |
| Median | XX.X |
| Max | xx.x |
| <=65 years | xxx ( xx.x) |
| >65 years | xxx ( xx.x) |
| Gender - n (%) | |
| Male | xxx ( xx.x) |
| Female | xxx ( xx.x) |
| Ethnicity - n (%) | |
| Hispanic or Latino | xxx ( xx.x) |
| Not Hispanic or Latino | xxx ( xx.x) |
| Race - n (%) | |
| Black or African American | xxx ( xx.x) |
| White | xxx ( xx.x) |
| Asian | xxx ( xx.x) |
| Native Hawaiian or Pacific Islander | xxx ( xx.x) |
| American-Indian or Alaska Native | xxx (xx.x) |
| Other | xxx (xx.x) |

PROGRAM\OUTPUT: T\_DEMOG.SAS\T\_DEMOG1.LST DATE(TIME): DDMMMYY(HH:MM)

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

#### Table 14.1.2

# Summary of Demographics (Population: Safety Evaluable Subjects)

| | Treatment Group |
|-----------------------------------|-----------------|
| | Ruxolitinib |
| Variable | (N=xxx) |
| Height at Screening (cm) | |
| n | XXX |
| Mean | xx.x |
| STD | X.XX |
| Min | xx.x |
| Median | xx.x |
| Max | xx.x |
| Height of Males at Screening (cm) | |
| n | XXX |
| Mean | xx.x |
| STD | x.xx |
| Min | XX.X |
| Median | xx.x |
| Max | XX.X |
| Height of Females at Screening ( | m) |
| n | xxx |
| Mean | XX.X |
| STD | X.XX |
| Min | XX.X |
| Median | XX.X |

PROGRAM\OUTPUT: T\_DEMOG.SAS\T\_DEMOG1.LST DATE(TIME): DDMMMYY(HH:MM)

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

#### Table 14.1.2

### Summary of Demographics (Population: Safety Evaluable Subjects)

| | Treatment Group |
|-------------------------------------|-----------------|
| | Ruxolitinib |
| Variable | (N=xxx) |
| Weight at Screening (kg) | |
| n | xxx |
| Mean | xx.x |
| STD | x.xx |
| Min | xx.x |
| Median | XX.X |
| Max | xx.x |
| Weight of Males at Screening (kg) | |
| n | XXX |
| Mean | xx.x |
| STD | x.xx |
| Min | xx.x |
| Median | xx.x |
| Max | xx.x |
| Weight of Females at Screening (kg) | |
| n | xxx |
| Mean | XX.X |
| STD | X.XX |
| Min | xx.x |
| Median | XX.X |
| Max | xx.x |

PROGRAM\OUTPUT: T\_DEMOG.SAS\T\_DEMOG1.LST DATE(TIME): DDMMMYY(HH:MM)

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

#### Table 14.1.2

### Summary of Demographics (Population: Safety Evaluable Subjects)

Treatment Group Ruxolitinib Variable (N=xxx)BMI  $(kg/m^2)$ n XXX Mean XX.X STD X.XX Min XX.X Median XX.X Max XX.X Resting Systolic Blood Pressure at Screening (mmHg) XXX Mean XX.X STD X.XX Min XX.X Median XX.X Max XX.X Resting Diastolic Blood Pressure at Screening (mmHg) n XXX Mean XX.X STD X.XX Min XX.X Median XX.X Max XX.X

PROGRAM\OUTPUT: T\_DEMOG.SAS\T\_DEMOG1.LST DATE(TIME): DDMMMYY(HH:MM)

### Incyte Corporation INCB 18424-258

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.3

Summary of Baseline Characteristics (Population: Safety Evaluable Subjects)

\_\_\_\_\_\_

Footnote Page

PROGRAM\OUTPUT: T DEMOG.SAS\T DISEASE1.LST

DATE(TIME): DDMMMYY(HH:MM)

Note: Baseline = the last measurement prior to 1st dose of study medication.

[1] Year since initial diagnosis = (first dose date - diagnosis date + 1)/365.25.

In case of partial date, first month of the year and/or first day of the month were used where applicable.

[2] ECOG Status: 0=Fully active, able to carry on all pre-disease performance without restriction

1=Restricted in physically strenuous activity but ambulatory and able to carry out

work of a light or sedentary nature

2=Ambulatory and capable of all selfcare but unable to carry out any work activities

Up and about more than 50% of waking hours

3=Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours

4=Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair

5=Dead

Reference: Listings 16.2.4.1 and 16.2.4.2.2

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

#### Table 14.1.3

Summary of Baseline Characteristics (Population: Safety Evaluable Subjects)

| Variable | Ruxolitinib<br>(N=xxx) |
|--------------------------------------------------|------------------------|
| variable | (N AAA) |
| Tumor Type - n (%) | |
| Primary Myelofibrosis | xxx ( xx.x) |
| Post Polycythemia Vera Myelofibrosis | xxx ( xx.x) |
| Post Essential Thrombocythemia Myelofibrosis | xxx ( xx.x |
| Time (year) Since Initial Diagnosis [1] | |
| n | XXX |
| Mean | x.x |
| STD | x.xx |
| Min | x.x |
| Median | <b>x.</b> x |
| Max | xx.x |
| With History Blood Component Transfusion - n (%) | |
| Yes | xxx ( xx.x) |
| Previous Hydroxyurea Use (HU) - n (%) | |
| Yes | xxx ( xx.x) |

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.3

Summary of Baseline Characteristics (Population: Safety Evaluable Subjects)

| Variable | Ruxolitinib<br>(N=xxx) |
|----------------------------------------|------------------------|
| Fibrosis Grade at Baseline - n (%) [2] | |
| 0 | xxx ( xx.x) |
| 1 | xxx ( xx.x) |
| 2 | xxx ( xx.x) |
| 3 | xxx ( xx.x) |
| Platelets at Baseline (GI/L) | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | XXX.X |
| Hemoglobin at Baseline (G/L) | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | xxx.x |

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.3

Summary of Baseline Characteristics (Population: Safety Evaluable Subjects)

| | Ruxolitinib |
|----------------------------------------|-------------|
| Variable | (N=xxx) |
| Neutrophils at Baseline (GI/L) | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | xxx.x |
| Leukocytes at Baseline (GI/L) | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | xxx.x |
| Total Cholesterol at Baseline (MMOL/L) | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | XXX.X |

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.3

Summary of Baseline Characteristics (Population: Safety Evaluable Subjects)

| | Ruxolitinib |
|---------------------------------------------|-------------|
| Variable | (N=xxx) |
| Creatinine at Baseline (UMOL/L) | |
| n | XXX |
| Mean | xxx.x |
| STD | XXX.XX |
| Min | xx.x |
| Median | XXX.X |
| Max | XXX.X |
| Aspartate Aminotransferase at Baseline (U/I | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | xxx.x |
| Alanine Aminotransferase at Baseline (U/L) | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | XXX.X |

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.3

Summary of Baseline Characteristics (Population: Safety Evaluable Subjects)

| | Ruxolitinib |
|--------------------------------|-------------|
| Variable | (N=xxx) |
| Bilirubin at Baseline (UMOL/L) | |
| n | XXX |
| Mean | XXX.X |
| STD | xxx.xx |
| Min | XX.X |
| Median | XXX.X |
| Max | XXX.X |
| Calcium at Baseline (MMOL/L) | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | xx.x |
| Median | XXX.X |
| Max | XXX.X |
| Glucose at Baseline (MMOL/L) | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | xxx.x |

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.3

Summary of Baseline Characteristics (Population: Safety Evaluable Subjects)

| | Ruxolitinib<br>(N=xxx) |
|--------------------------------|------------------------|
| Variable | |
| Potassium at Baseline (MMOL/L) | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | XXX.X |
| Sodium at Baseline (MMOL/L) | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | xxx.x |
| DIPSS Score | |
| HIGH RISK (5-6) | xxx ( xx.x) |
| INTERMEDIATE-2 (3-4) | xxx (xx.x) |

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.3

Summary of Baseline Characteristics (Population: Safety Evaluable Subjects)

| | Ruxolitinib |
|------------------------------------------|-------------|
| Variable | (N=xxx) |
| Spleen Volume at Baseline (cm^3) | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | XXX.X |
| Spleen Palpation Length at Baseline (cm) | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | XXX.X |
| Total Symptom Score at Baseline | |
| n | XXX |
| Mean | XXX.X |
| STD | XXX.XX |
| Min | XX.X |
| Median | XXX.X |
| Max | xxx.x |

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.3

Summary of Baseline Characteristics (Population: Safety Evaluable Subjects)

| Variable | Ruxolitinib<br>(N=xxx) |
|----------------------|------------------------|
| ECOG at Baseline [3] | |
| 0 | xxx ( xx.x) |
| 1 | xxx ( xx.x) |
| 2 | xxx ( xx.x) |
| 3 | xxx ( xx.x) |
| 4 | xxx ( xx.x) |
| Percent at Baseline | |
| Yes | xxx ( xx.x) |
| No | xxx ( xx.x) |
| Missing | xxx ( xx.x) |

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

#### Table 14.1.4

Summary of Medical History by MedDRA System Organ Class and Preferred Term (Population: Safety Evaluable Subjects)

| MedDRA System Organ Class<br>Preferred Term | Ruxolitinib<br>(N=xxx) |
|---------------------------------------------|------------------------|
| Subjects With Any Medical History | xxx (xxx.x) |
| SOC 1 | xxx (xxx.x) |
| Preferred Term 1 | xxx (xxx.x) |

PROGRAM\OUTPUT: T\_xxxxx.SAS\T\_xxxxxx.LST DATE(TIME): DDMMMYY(HH:MM)

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.5.1

# Summary of Prior Medications (Population: Safety Evaluable Subjects)

| ATC Class/WHO Preferred Term | Ruxolitinib<br>(N=xxx) |
|-----------------------------------------|------------------------|
| <br>Subjects With Any Prior Medications | xxx (xxx.x) |
| WHO Drug Class 1 | xxx (xxx.x) |
| WHO Preferred Term 1 | xxx (xxx.x) |
| WHO Preferred Term 2 | xxx (xxx.x) |
| WHO Preferred Term 3 | xxx (xxx.x) |
| WHO Preferred Term 4 | xxx (xxx.x) |
| WHO Drug Class 2 | xxx (xxx.x) |
| WHO Preferred Term 1 | xxx (xxx.x) |
| WHO Preferred Term 2 | xxx (xxx.x) |
| WHO Preferred Term 3 | xxx (xxx.x) |
| WHO Preferred Term 4 | xxx (xxx.x) |

PROGRAM\OUTPUT: T\_DEMOG.SAS\T\_DEMOG1.LST DATE(TIME): DDMMMYY(HH:MM)

Incyte Corporation
INCB 18424-258
Statistical Analysis Plan - Final
17 JAN 2012


DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.5.2

Summary of Concomitant Medications (Population: Safety Evaluable Subjects)

NOTE TO THE PROGRAMMER: THIS TABLE WILL BE SIMILARLY PROGRAMMED AS Table 14.1.5.1

Incyte Corporation
INCB 18424-258
Statistical Analysis Plan - Final
17 JAN 2012


DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.5.3

Summary of Prior Anti-Cancer Treatment (Population: Safety Evaluable Subjects)

NOTE TO THE PROGRAMMER: THIS TABLE WILL BE SIMILARLY PROGRAMMED AS Table 14.1.5.1

71

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.6.1

Summary of Change in Status of Blood Component Transfusion Dependency by Baseline Platelet Count Group (Population: Safety Evaluable Subjects)

| Pattern of Change in | | Baseline Pla | | |
|---|---|---|---|---|
| Dependency | Time | 50-75 GI/L | >75 GI/L | Total |
| Status | Interval | N n (%) | N n (%) | N n (%) |
| Depend. to Indep. | 8 Weeks before Day 1 to Final 8 Weeks | xx xx(xx.x) | xx xx (xx.x) | xx xx (xx.x) |
| | 12 Weeks before Day 1 to Final 12 Weeks | xx xx(xx.x) | xx xx (xx.x) | xx xx (xx.x) |
| Indep. to Depend. | 8 Weeks before Day 1 to Final 8 Weeks<br>12 Weeks before Day 1 to Final 12 Weeks | xx xx(xx.x)<br>xx xx(xx.x) | xx xx (xx.x)<br>xx xx (xx.x) | xx xx (xx.x)<br>xx xx (xx.x) |

PROGRAM\OUTPUT: T xxxxx.SAS\T xxxx.LST

DATE (TIME): ddmmmyyyy (hh:mm)

Note 1: N = # subjects at the beginning of the first interval, and n (%) = # (%) subjects at the end of the second interval. The first interval covered within 8 (or 12) weeks prior to Day 1, and the second interval covered last 8 (or 12) weeks after Day 1. Percents are calculated as n/N\*100 for each row of each group.

Note 2: Transfusion dependence is defined as subjects received at least 1 unit of red blood cell product(s) during the given period. Independence is defined as subjects received 0 unit of red blood cell product(s) during the given period.

Reference: xxxx
DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.1.6.2

Summary of Blood Component Transfusions by Baseline Platelet Count Group (Population: Safety Evaluable Subjects)

| | Baseline Pla | | |
|---|---|---|---|
| | 50-75 GI/L | > 75 GI/L | <br>Total |
| Variable | (N = xx) | (N = xx) | (N = xx) |
| Monthly Units of RBC Transfusion: Baseline | | | |
| n | | | |
| Mean (Std) | | | |
| Median | | | |
| Min, Max | | | |
| Total Units of RBC Transfusion: Post-Baseline | | | |
| n | | | |
| Mean (Std) | | | |
| Median | | | |
| Min, Max | | | |
| Monthly Units of RBC Transfusion: Post-Baseline | | | |
| n | | | |
| Mean (Std) | | | |
| Median | | | |
| Min, Max | | | |
| PROGRAM\OUTPUT: T xxxxx.SAS\T xxxx.LST | | DATE(TIME): d | dmmmyyyy(hh:mm |

PROGRAM\OUTPUT: T\_XXXXX.SAS\T\_XXXX.LST

Note 1: Total units = all units during the treatment phase from Day 1 to the last scheduled visit. Note 2: Monthly units = total units divided by the treatment duration (in months where 1 month = 30.4375 days). Reference: Listing xxxxx.

DATE (TIME): DDMMMYY (HH:MM)

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

## Table 14.2.1.1

Summary of Correlation of Final Titrated Dose vs. Percent Change from Baseline in Spleen Volume at Week 24 and vs. Percent Change in Total Symptom Score at Week 24 (Population: ITT Subjects)

| | Ruxolitinib |
|---|---|
| Variable | (N=xxx) |
| Dose vs. % Chg in Spleen Volume | |
| Sample size, n | XXX |
| Pearson correlation coefficient - raw value | X.XXX |
| p-value from t-test | 0.xxx |
| Estimated corr coeff - Fisher transformation (95% CI) | x.xxx (x.xxx, x.xxx) |
| Dose vs. % Chg in Total Symptom Score | |
| Sample size, n | XXX |
| Pearson correlation coefficient - raw value | X.XXX |
| p-value from t-test | 0.xxx |
| Estimated corr coeff - Fisher transformation (95% CI) | x.xxx (x.xxx, x.xxx) |

PROGRAM\OUTPUT: T xxxxx.SAS\T xxxxxx.LST

Note: t-test was based on the raw Pearson correlation coefficient; and 95% confidence interval is based on the Approximation from Fisher's r-to-z transformation.

Reference: Listings 16.2.6.

NOTE TO THE TEAM: if protocol is further amended, we should consistently specify p-value and 95% CI calculation, that they all come from Fisher r-to-z transformation.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.2.1.2

Summary of Correlation of Final Titrated Dose vs. Percent Change from Baseline in Spleen Volume at Week 24 and vs. Percent Change in Total Symptom Score at Week 24: Sensitivity Analysis 1 (Population: Per-Protocol Subjects)

NOTE TO THE PROGRAMMER: this table will be similarly programmed as 14.2.1.1.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.2.1.3

Summary of Correlation of Final Titrated Dose vs. Percent Change from Baseline in Spleen Volume at Week 24 and vs. Percent Change in Total Symptom Score at Week 24: Sensitivity Analysis 2 (Population: ITT Subjects)

NOTE TO THE PROGRAMMER: this table will be similarly programmed as 14.2.1.1.

• Footnote need to add MI model and procedure for this sensitivity analysis.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.2.2.1

Summary of Spleen Volume (cm^3) by Study Week and Final Titrated Dose Group (Population: ITT Subjects)

| | | Ru | xolitinib Final Ti | trated Dose (mg) Gr | roup |
|---|---|---|---|---|---|
| Study Week<br>Variable | Total (N=xxx) | < 5<br>(N=xx) | >5 to 15<br>(N=xx) | >15 to 25<br>(N=xx) | >25<br>(N=xx) |
| Baseline | | | | | |
| n | xxx | xx | XX | XX | XX |
| Mean | xxxx.x | xxxx.x | xxxx.x | XXXX.X | xxxx.x |
| Std | xxxx.xx | xxxx.xx | xxxx.xx | xxxx.xx | xxxx.xx |
| Median | XXXX.X | xxxxx.x | xxxx.x | xxxx.x | xxxx.x |
| Min, Max | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) |
| Week 24: raw | | | | | |
| n | xxx | xx | xx | XX | XX |
| Mean | xxxx.x | xxxx.x | xxxx.x | XXXX.X | XXXX.X |
| Std | xxxx.xx | xxxx.xx | xxxx.xx | XXXX.XX | xxxx.xx |
| Median | xxxx.x | xxxxx.x | xxxx.x | xxxx.x | xxxx.x |
| Min, Max | (xxxx.x, xxxx.x | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) |

PROGRAM\OUTPUT: T\_XXXXX.SAS\T\_XXXXXX.LST DATE(TIME): DDMMMYY(HH:MM)

Reference: Listing 16.2.6.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.2.2.1

Summary of Spleen Volume (cm^3) by Study Week and Final Titrated Dose Group (Population: ITT Subjects)

| | | Rux | colitinib Final Tit | rated Dose (mg) Gr | oup |
|---|---|---|---|---|---|
| Study Week<br>Variable | Total<br>(N=xxx) | < 5<br>(N=xx) | >5 to 15<br>(N=xx) | >15 to 25<br>(N=xx) | >25<br>(N=xx) |
| Week 24: Chg from Baseline | | | | | |
| n | XXX | XX | XX | XX | XX |
| Mean | xxxx.x | xxxx.x | xxxx.x | xxxx.x | xxxx.x |
| Std | xxxx.xx | xxxx.xx | xxxx.xx | xxxx.xx | xxxx.xx |
| Median | xxxx.x | xxxxx.x | xxxx.x | xxxx.x | xxxx.x |
| Min, Max | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) |
| p-value from t-test | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx |
| p-value from WRS-test | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx |
| Week 24: %Chg from Baseline | 2 | | | | |
| n | xxx | xx | xx | xx | xx |
| Mean | xxxx.x | xxxx.x | xxxx.x | xxxx.x | xxxx.x |
| Std | xxxx.xx | xxxx.xx | xxxx.xx | xxxx.xx | xxxx.xx |
| Median | xxxx.x | xxxxx.x | xxxx.x | xxxx.x | xxxx.x |
| Min, Max | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) |
| p-value from t-test | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx |
| p-value from WRS-test | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx |

PROGRAM\OUTPUT: T\_xxxxx.SAS\T\_xxxxxx.LST DATE(TIME): DDMMMYY(HH:MM)

Reference: Listing 16.2.6.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.2.2.2

Summary of Proportion of Subjects with >= 35% Reduction from Baseline in Spleen Volume at Week 24 by Final Titrated Dose Group (Population: ITT Subjects)

| Study Week<br>Variable | Total (N=xxx) | < 5<br>(N=xx) | >5 to 15<br>(N=xx) | >15 to 25<br>(N=xx) | >25<br>(N=xx) |
|---|---|---|---|---|---|
| Week 24: Reduction of >= 35% | | | | | |
| No | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Yes | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 95% CI for response rate [1] | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Reasons for not Achieving The reduction of >= 35% - n (%) | | | | | |
| Discontinued prior to Week 24 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Data missing/out of window | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

PROGRAM\OUTPUT: T\_XXXXX.SAS\T\_XXXXXX.LST DATE(TIME): DDMMMYY(HH:MM)

[1]: 95% CI is from exact binomial distribution.

Reference: Listing 16.2.6.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.2.2.3

Summary of Proportion of Subjects with >= 10% Reduction from Baseline in Spleen Volume at Week 24 by Final Titrated Dose Group (Population: ITT Subjects)

NOTE TO THE PROGRAMMER: this table will be programmed similarly to Table 14.2.2.2.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.2.3.1

Summary of Total Symptom Score by Study Week and Final Titrated Dose Group (Population: ITT Subjects)

NOTE TO THE PROGRAMMER: this table will be programmed similarly to Table 14.2.2.1 but Study Weeks will be 0, 4, 8, 12, 16, 20, 24.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.2.3.2

Summary of Proportion of Subjects with >= 50% Reduction from Baseline in Total Symptom Score by Study Week and Final Titrated Dose Group (Population: ITT Subjects)

NOTE TO THE PROGRAMMER: this table will be similarly program as Table 14.2.2.2 but will not derive/display reason of not achieving a response.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

NOTE TO THE PROGRAMMER: this table will be similarly program as Table 14.2.2.2 but will not derive/display reason of not achieving a response.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.2.4.1

Summary of Spleen Palpation Length Data by Study Week and Final Titrated Dose Group (Population: ITT Subjects)

NOTE TO THE PROGRAMMER: this table will be programmed similarly to Table 14.2.2.1 but Study Weeks will be the nominal weeks where spleen length data are scheduled to be collected.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.2.4.2

Summary of Proportion of Subjects with >= 50% Reduction from Baseline in Spleen Palpation Length by Study Week and Final Titrated Dose Group (Population: ITT Subjects)

NOTE TO THE PROGRAMMER: this table will be similarly program as Table 14.2.2.2 but will not derive/display reason of not achieving a response.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.2.4.3

Summary of Proportion of Subjects with >= 20% Reduction from Baseline in Spleen Palpation Length by Study Week and Final Titrated Dose Group (Population: ITT Subjects)

NOTE TO THE PROGRAMMER: this table will be similarly program as Table 14.2.2.2 but will not derive/display reason of not achieving a response.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.2.5.1

Summary of Patient Global Impression of Change Score by Study Week and Final Titrated Dose Group (Population: ITT Subjects)

NOTE TO THE PROGRAMMER: this table will be similarly program as Table 14.2.2.1 but no change and percent change will be derived.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

NOTE TO THE PROGRAMMER: this table will be similarly program as Table 14.2.2.1.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

NOTE TO THE PROGRAMMER: this table will be similarly program as Table 14.2.2.1.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.3.1.1

Summary of Exposure and Duration of Exposure to Study Medication Through Week 24 by Final Titrate Dose Level (Population: Safety Evaluable Subjects)

| | Ruxolitinib Final Titrated Dose (mg) | | | | |
|---|---|---|---|---|---|
| Variable | Total<br>(N=xxx) | < 5<br>(N=xx) | >5 to 15<br>(N=xx) | >15 to 25<br>(N=xx) | >25<br>(N=xx) |
| Duration of Treatment (weeks) [1] | | | | | |
| n | XXX | XX | XX | XX | xx |
| Mean | XXXX.X | XXXX.X | XXXX.X | XXXX.X | xxxx.x |
| Std | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| Median | XXXX.X | XXXXX.X | XXXX.X | XXXX.X | xxxx.x |
| Min, Max | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| <=30 Days | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 31-90 Days | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 91-120 Days | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 121-150 Days | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >150 Days | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patient Year [2] | X.XX | x.xx | x.xx | x.xx | x.xx |

PROGRAM\OUTPUT: T xxxx.SAS\T xxxx.LST

DATE(TIME): ddmmmyy(hh:mm)

Reference: Listing 16.2.7.1.1.

<sup>[1]</sup> Duration of treatment is calculated as (last dose date during the treatment period - first dose date +1)/7 disregard interruptions in between.

<sup>[2]</sup> Patient year is calculated based on duration of treatment.

<sup>[3]</sup> Average daily dose is calculated as total dose (mg) divided by duration of treatment expressed in days.

<sup>[4]</sup> Overall compliance is calculated as (total # of tablets consumed)/(total # of tablets expected to be consumed)\*100, where total # of tablets expected to be consumed is based on prescribed doses (including interruption) from CRF domain of EX.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.3.1.1

Summary of Exposure and Duration of Exposure to Study Medication Through Week 24 by Final Titrate Dose Level (Population: Safety Evaluable Subjects)

| | Ruxolitinib Final Titrated Dose (mg) | | | | |
|---|---|---|---|---|---|
| Variable | Total<br>(N=xxx) | < 5<br>(N=xx) | >5 to 15<br>(N=xx) | >15 to 25<br>(N=xx) | >25<br>(N=xx) |
| Average Daily Dose (mg) [3] | | | | | |
| n | XXX | XX | XX | XX | XX |
| Mean | XXXX.X | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| Std | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| Median | XXXX.X | XXXXX.X | XXXX.X | XXXX.X | XXXX.X |
| Min, Max | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Last 7 Days Average Daily Dose (mg) | | | | | |
| n | XXX | XX | XX | XX | XX |
| Mean | XXXX.X | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| Std | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| Median | XXXX.X | XXXXX.X | XXXX.X | XXXX.X | XXXX.X |
| Min, Max | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |

PROGRAM\OUTPUT: T xxxx.SAS\T xxxx.LST

DATE(TIME): ddmmmyy(hh:mm)

- [1] Duration of treatment is calculated as (last dose date during the treatment period first dose date +1)/7 disregard interruptions in between.
- [2] Patient year is calculated based on duration of treatment.
- [3] Average daily dose is calculated as total dose (mg) divided by duration of treatment expressed in days.
- [4] Overall compliance is calculated as (total # of tablets consumed)/(total # of tablets expected to be consumed)\*100, where total # of tablets expected to be consumed is based on prescribed doses (including interruption) from CRF domain of EX.

Reference: Listing 16.2.7.1.1.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.3.1.1

Summary of Exposure and Duration of Exposure to Study Medication Through Week 24 by Final Titrate Dose Level (Population: Safety Evaluable Subjects)

| | | Rux | colitinib Final | Titrated Dose ( | mg) |
|---|---|---|---|---|---|
| Variable | Total<br>(N=xxx) | < 5<br>(N=xx) | >5 to 15<br>(N=xx) | >15 to 25<br>(N=xx) | >25<br>(N=xx) |
| Overall Compliance (%) [4] | | | | | |
| <=50 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >51-80 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >80 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

PROGRAM\OUTPUT: T xxxx.SAS\T xxxx.LST

DATE(TIME): ddmmmyy(hh:mm)

- [1] Duration of treatment is calculated as (last dose date during the treatment period first dose date +1)/7 disregard interruptions in between.
- [2] Patient year is calculated based on duration of treatment.
- [3] Average daily dose is calculated as total dose (mg) divided by duration of treatment expressed in days.
- [4] Overall compliance is calculated as (total # of tablets consumed)/(total # of tablets expected to be consumed)\*100, where total # of tablets expected to be consumed is based on prescribed doses (including interruption) from CRF domain of EX.

Reference: Listing 16.2.7.1.1.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.3.1.2

Summary of Exposure and Duration of Exposure to Study Medication Through Week 4 by Final Titrate Dose Level (Population: Safety Evaluable Subjects)

NOTE TO THE PROGRAMMER: this table will programmed similarly to Table 14.3.1.1 but present only average daily dose.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.3.1.3

Summary of Average Daily Dose of Ruxolitinib by Study Week and Final Titrate Dose Level (Population: Safety Evaluable Subjects)

| | | Ruxolitinib Final Titrated Dose (mg) | | | |
|---|---|---|---|---|---|
| <i>J</i> ariable | Total<br>(N=xxx) | < 5<br>(N=xx) | >5 to 15<br>(N=xx) | >15 to 25<br>(N=xx) | >25<br>(N=xx) |
| Average Daily Dose (mg) for Week | 1 | | | | |
| n | xxx | XX | XX | XX | XX |
| Mean | xxxx.x | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| Std | xxxx.xx | XXXX.XX | XXXX.XX | XXXX.XX | xxxx.xx |
| Median | xxxx.x | XXXXX.X | XXXX.X | XXXX.X | xxxx.x |
| Min, Max | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |

Average Daily Dose (mg) for Week 2 . . .

PROGRAM\OUTPUT: T xxxx.SAS\T xxxx.LST

DATE(TIME): ddmmmyy(hh:mm)

Reference: Listing 16.2.7.1.1.

NOTE TO THE PROGRAMMER: Table is continued to Week 48 as long as data is available.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.3.2.1

Overall Summary of Treatment-Emergent Adverse Events by Dose Ever Received (Population: Safety Evaluable Subjects)

| | All | Do | se Level (mg | () Subjects | Ever Recei | Lved |
|---|---|---|---|---|---|---|
| Variable | Subjects<br>(N=23) | <=5<br>(N=2) | >5 10<br>(N=23) | >10 15<br>(N=14) | >15 20<br>(N=7) | >20 25<br>(N=1) |
| Treatment-Emergent Adverse Events (TEAE) Reported | 33 | 1 | 8 | 21 | 3 | 0 ( 0.0) |
| Subjects with a TEAE | 10 ( 43.5) | 1 (50.0) | 3 (13.0) | 5 ( 35.7) | 1 (14.3) | 0 ( 0.0) |
| Subjects with a Treatment-Related TEAE | 2 ( 8.7) | 0 ( 0.0) | 1 ( 4.3) | 1 ( 7.1) | 0 ( 0.0) | 0 ( 0.0) |
| Subjects with a Serious TEAE | 2 ( 8.7) | 1 (50.0) | 0 ( 0.0) | 1 ( 7.1) | 0 ( 0.0) | 0 ( 0.0) |
| Subjects with TEAE of Grade 3 or Higher | 4 ( 17.4) | 1 (50.0) | 1 ( 4.3) | 2 ( 14.3) | 0 ( 0.0) | 0 ( 0.0) |
| Subjects with a Dose Increase Due to TEAE | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) |
| Subjects with a Dose Reduction Due to TEAE | 1 ( 4.3) | 0 ( 0.0) | 0 ( 0.0) | 1 ( 7.1) | 0 ( 0.0) | 0 ( 0.0) |
| Subjects with Procedures Performed Due to TEAE | 2 ( 8.7) | 0 ( 0.0) | 0 ( 0.0) | 2 (14.3) | 0 ( 0.0) | 0 ( 0.0) |
| Subjects with a TEAE requiring Concomitant Medication | 5 ( 21.7) | 0 ( 0.0) | 1 ( 4.3) | 4 (28.6) | 0 ( 0.0) | 0 ( 0.0) |
| Subjects with Study Drug Withdrawn Due to TEAE | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) |
| Subjects with an TEAE Leading to Discontinuation from the Study | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) |
| Subjects with a TEAE Leading to Death | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) | 0 ( 0.0) |

PROGRAM\OUTPUT: T AESUM1.SAS\T AE1.LST

DATE (TIME): 12DEC11(11:30)

Note 1:TEAEs: AEs that began or worsened from baseline following the first administration of the study drug.

Note 2:Treatment-Related AEs:TEAEs with a possible, probable, definite, or missing casuality.

Note 3:Severity vs CTCAE Grade: Mild=Grade 1, Moderate=Grade 2, Severe=Grade 3, Life-Threatening=Grade 4.

Note 4:For an AE that occurred for more than once to a subject, it is counted in the lowest dose when the highest severity grade is recorded.

Reference: Listings 16.2.7.2.1

NOTE to the reviewer: numbers in the shell is from draft DMC output and is intended to show shell only.

Incyte Corporation Statistical Analysis Plan - Final INCB 18424-258 Statistical Analysis Plan - Final 17 JAN 2012

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: First DMC-Draft

Table 14.3.2.2.1

Summary of Subjects Reporting Treatment-Emergent Adverse Events (All Causalities) by MedDRA System Organ Class, Preferred Term, and Maximum Severity (Population: Safety Evaluable Subjects)

NOTE TO THE PROGRAMMER: shell will following the standard output.

• Reference: 16.2.7.2.1

DATE (TIME): 12DEC11(11:30)

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: First DMC-Draft

Table 14.3.2.2.2

Summary of Subjects Reporting Treatment-Emergent Adverse Events (All Causalities) by
MedDRA System Organ Class, Preferred Term, and Dose Level Ever Received
(Population: Safety Evaluable Subjects)

| | CTCAE Grade | | | | | |
|---|---|---|---|---|---|---|
| Variable | All<br>Subjects<br>(N=23) | 0<br>(N=2) | >5 10<br>(N=23) | >10 15<br>(N=14) | >15 20<br>(N=7) | >20 25<br>(N=1) |
| Number (%) of Subjects With Any TEAEs | 10 ( 43.5) | 1 (50.0) | 3 (13.0) | 5 ( 35.7) | 1 ( 14.3) | 0 ( 0.0) |
| Blood and lymphatic system disorders | 1 (4.3) | 0 (0.0) | 0 (0.0) | 1 (7.1) | 0 (0.0) | 0 ( 0.0) |
| Anaemia | 1 (4.3) | 0 (0.0) | 0 (0.0) | 1 (7.1) | 0 (0.0) | 0 ( 0.0) |
| Gastrointestinal disorders | 6 ( 26.1) | 0 (0.0) | 0 (0.0) | 4 ( 28.6) | 2 ( 28.6) | 0 ( 0.0) |
| Abdominal pain | 2 (8.7) | 0 (0.0) | 1 (4.3) | 1 (7.1) | 0 (0.0) | 0 ( 0.0) |
| Anorectal discomfort | 1 (4.3) | 0 (0.0) | 0 (0.0) | 1 (7.1) | 0 (0.0) | 0 ( 0.0) |
| Diarrhoea | 3 (13.0) | 0 (0.0) | 0 (0.0) | 2 (14.3) | 1 (14.3) | 0 ( 0.0) |
| Dry mouth | 1 (4.3) | 0 (0.0) | 0 (0.0) | 0 (0.0) | 1 (14.3) | 0 ( 0.0) |
| Haemorrhoidal haemorrhage | 1 (4.3) | 0 (0.0) | 0 (0.0) | 1 (7.1) | 0 (0.0) | 0 ( 0.0) |
| Nausea | 1 (4.3) | 0 (0.0) | 0 (0.0) | 1 (7.1) | 0 (0.0) | 0 (0.0) |

PROGRAM\OUTPUT: T AESUM1.SAS\T AE2.LST

Note 1:TEAEs: AEs that began or worsened from baseline following the first administration of the study drug.

Note 2:N=the number of subjects who ever took a dose within the dose group, based on which the percent is calculated.

Note 3:For an AE that occurred for more than once to a subject, it is counted in the lowest dose when

the highest severity grade is recorded.

Reference: Listings 16.2.7.2.1

NOTE to the reviewer: numbers in the shell is from draft DMC output and is intended to show shell only.

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: First DMC-Draft

Table 14.3.2.3.1

Summary of Subjects Reporting Treatment-Emergent Adverse Events (All Causalities) by

MedDRA Preferred Term (Sorted by Decreasing Frequency) and Maximal Severity

(Population: Safety Evaluable Subjects)

NOTE TO THE PROGRAMMER: shell will following the standard output.

• Reference: 16.2.7.2.1

**Incyte Corporation** 

INCB 18424-258

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: First DMC-Draft

Table 14.3.2.3.2

Summary of Subjects Reporting Treatment-Emergent Adverse Events (All Causalities) by

MedDRA Preferred Term (Sorted by Decreasing Frequency) and Dose Ever Received

(Population: Safety Evaluable Subjects)

NOTE TO THE PROGRAMMER: shell will following the standard output and table will be similarly programmed as 14.3.2.2.2.

• Reference: 16.2.7.2.1

NOTE: Shells for the following tables are not provided here but they will be programmed similarly to those presented above.

| 14.3.2.3.2 | Summary of Subjects Reporting Treatment-Emergent Adverse<br>Events (All Causalities) by MedDRA Preferred Term (Sorted by<br>Decreasing Frequency) and Dose Level Ever Received | Safety |
|---|---|---|
| 14.3.2.3.3 | Summary of Subjects Reporting Treatment-Emergent Hemorrhage<br>Adverse Events (All Causalities) by MedDRA Preferred Term and<br>Dose Level Ever Received | Safety |
| 14.3.2.3.4 | Summary of Subjects Reporting Treatment-Emergent Hemorrhage<br>Adverse Events (All Causalities) of Grade 3 or Higher by MedDRA<br>Preferred Term and Dose Level Ever Received | Safety |
| 14.3.2.4.1 | Summary of Subjects Reporting Treatment-Emergent Treatment-Related Adverse Events (All Causalities) by MedDRA System Organ Class, Preferred Term, and Maximum Severity | Safety |
| 14.3.2.4.2 | Summary of Subjects Reporting Treatment-Emergent Treatment-Related Adverse Events (All Causalities) by MedDRA System Organ Class, Preferred Term, and Dose Level Ever Received | Safety |
| 14.3.2.5.1 | Summary of Subjects Reporting Treatment-Emergent Serious<br>Adverse Events (All Causalities) by MedDRA System Organ Class,<br>Preferred Term, and Dose Level Ever Received | Safety |
| 14.3.2.6 | Summary of Subjects Reporting Treatment-Emergent Adverse Events (All Causalities) Leading to Study Medication Decrease or Interruption by MedDRA System Organ Class, Preferred Term, and Dose Level Ever Received | Safety |
| 14.3.2.7 | Summary of Subjects Reporting Treatment-Emergent Adverse<br>Events (All Causalities) Leading to Study Discontinuation by<br>MedDRA System Organ Class, Preferred Term, and Dose Level<br>Ever Received | Safety |
| 14.3.2.8 | Summary of Subjects Reporting Treatment-Emergent Adverse<br>Events (All Causalities) Leading to On-Study Death by MedDRA<br>System Organ Class, Preferred Term, and Dose Level Ever<br>Received | Safety |

NOTE: the following lab tables will be programmed according to standard output.

| 14.3.3.1.1 | Summary of Laboratory Values – Hematology | Safety |
|---|---|---|
| 14.3.3.1.2 | Shift Summary of Laboratory Values in Normal Ranges - | Safety |
| | Hematology | |
| 14.3.3.2.1 | Summary of Laboratory Values – Serum Chemistry | Safety |
| 14.3.3.2.2 | Shift Summary of Laboratory Values in Normal Ranges – Serum | Safety |
| | Chemistry | |
| 14.3.3.3.1 | Summary of Laboratory Values – Coagulation | Safety |
| 14.3.3.3.2 | Shift Summary of Laboratory Values in Normal Ranges – | Safety |
| | Coagulation | |
| 14.3.3.4.1 | Summary of Laboratory Values – Urinalysis | Safety |
| 14.3.3.4.2 | Shift Summary of Laboratory Values in Normal Ranges – Urinalysis | Safety |
| 14.3.3.5.1 | Shift Summary of Laboratory Values in CTC Grade - To the Worst | Safety |
| | Abnormal Value (Tests with One Directional CTC Grade) | |
| 14.3.3.5.2 | Shift Summary of Laboratory Values in CTC Grade - To the Worst | Safety |
| | Abnormal Value (Tests with Two Directional CTC Grade) | - |

DATE (TIME): DDMMMYY (HH:MM)

PROTOCOL: INCB 18424-258  VERSION: Final DRUG/INDICATION: Ruxolitinib/Myelofibrosis

Table 14.3.3.6.1

Summary of Subjects with Treatment Emergent Thrombocytopenia of Grade 4 as Derived from Laboratory Data by Last Dose Before Onset (Population: Safety Evaluable Subjects)

| | Dose Level (mg) Subjects Ever Received | | | | | | |
|---|---|---|---|---|---|---|---|
| | All<br>Subjects | <=5 | >5 10 | >10 15 | >15 20 | >20 25 | >25 |
| MedDRA Preferred Term | (N=xx) | N=xx | N=xx | N=xx | N=xx | N=XX | N=xx |
| Number (%) of Subjects With Grade 4 Thrombocytopenia [1] | xx ( xx.x) | xx xx% | XX XX% | XX XX% | XX XX% | xx xx% | XX XX% |

PROGRAM\OUTPUT: T xxxx.SAS\T xxxxx.LST

Treatment-Emergent AEs: AEs that began or worsened from baseline following the first administration of study drug. Note: Subjects are counted only once under in the lowest dose group.

Note: N=the number of subjects who ever took a dose within the dose group, based on which the percent is calculated. Note: AEs that occurred following the date of treatment crossover were not included.

[1] Grade 4 Thrombocytopenia is defined as any occurrence of a treatment emergent hematology lab below 25 GI/L Reference: Listing 16.2.8.1.4

DRUG/INDICATION: Ruxolitinib/Myelofibrosis VERSION: Final

Table 14.3.3.6.2

Summary of Subjects with Treatment Emergent Anemia of Grade 4 as Derived from Laboratory Data by Last Dose Before Onset
(Population: Safety Evaluable Subjects)

NOTE TO THE PROGRAMMER: similarly program this as Table 14.3.3.6.1, just need to update footnote about G4 anemia.

## Incyte Corporation INCB 18424-258

NOTE: the following vital sign tables will be programmed according to standard output.

| 14.3.4.1 | Summary of Systolic Blood Pressure | Safety |
|----------|-------------------------------------|--------|
| 14.3.4.2 | Summary of Diastolic Blood Pressure | Safety |
| 14.3.4.3 | Summary of Heart Rate | Safety |
| 14.3.4.4 | Summary of Respiratory Rate | Safety |
| 14.3.4.5 | Summary of Body Temperature | Safety |

NOTE: the following laboratory tables will be programmed according to standard output.

| 14.2.1.1 | Scatter Plot of Percent Change from Baseline in Spleen Volume at | ITT |
|---|---|---|
| | Week 24 vs. Final Titrated Dose Level | |
| 14.2.1.2 | Scatter Plot of Percent Change from Baseline in Total Symptom | ITT |
| | Score at Week 24 vs. Final Titrated Dose Level | |
| 14.2.1.3 | Scatter Plot of Percent Change from Baseline in Spleen Volume vs. | ITT |
| | Percent Change in Total Symptom Score at Week 24 | |
| 14.2.2.1 | Bar Plot of Percent of Subjects with >= 35% Reduction from | ITT |
| | Baseline in Spleen Volume at Week 24 by Final Titrated Dose | |
| | Group | |
| 14.2.2.2 | Bar Plot of Percent of Subjects with >= 10% Reduction from | ITT |
| | Baseline in Spleen Volume at Week 24 by Final Titrated Dose | |
| | Group | |
| 14.2.2.3.1 | Mean (95%) Percent Change from Baseline in Spleen Volume at | ITT |
| | Week 24 | |
| 14.2.2.3.2 | Mean (95%) Percent Change from Baseline in Spleen Volume at | ITT |
| | Week 24 by Final Titrated Dose Group | |
| 14.3.1.1.1 | Subject Laboratory Value over Time: Hemoglobin (G/L) | Safety |
| 14.3.1.1.2 | Mean (95% CI) Laboratory Value Over Time: Hemoglobin (G/L) | Safety |
| 14.3.1.2.1 | Subject Laboratory Value over Time: Platelet (GI/L) | Safety |
| 14.3.1.2.2 | Mean (95% CI) Laboratory Value Over Time: Platelet (GI/L) | Safety |
| 14.3.1.3.1 | Subject Laboratory Value over Time: WBC (GI/L) | Safety |
| 14.3.1.3.2 | Mean (95% CI) Laboratory Value Over Time: WBC (GI/L) | Safety |
| 14.3.1.4.1 | Subject Laboratory Value over Time: Neutrophils (GI/L) | Safety |
| 14.3.1.4.2 | Mean (95% CI) Laboratory Value Over Time: Neutrophils (GI/L) | Safety |